CLINICAL TRIAL: NCT00791258
Title: A Prospective, Open-Label, Titration Study to Evaluate the Efficacy and Safety Safety of AZOR in Multiple Subgroups of Hypertensive Subjects Who Are Non-Responders to Anti-Hypertensive Monotherapy
Brief Title: A Dose Escalation Study of a Combination Antihypertensive Drug in the Treatment of Various Groups of Patients Who do Not Respond to Single Drug Treatment of Their High Blood Pressure
Acronym: BP CRUSH
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Collaborators: Integrium (Industry)
Responsible Party: Diector of Medical Research and Strategy, Daiichi Sankyo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CS8663-404
Record Dates: First submitted 2008-11-13; First posted 2008-11-14 (Estimated); Results first posted 2010-09-29 (Estimated); Last update posted 2019-01-09 (Actual); Status verified 2010-09

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Amlodipine; Olmesartan Medoxomil; Amlodipine Besylate, Olmesartan Medoxomil Drug Combination; Hydrochlorothiazide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Azor tablets and hydrochlorothiazide tablets (if necessary) will be administered for up to 20 weeks
  Interventions: Drug: amlodipine and olmesartan medoxomil tablets; Drug: hydrochlorothiazide tablets

INTERVENTIONS:
Drug: amlodipine and olmesartan medoxomil tablets — amlodipine and olmesartan medoxomil tablets administered orally, once daily for up to 20 weeks
  Other Names: AZOR Tablets
Drug: hydrochlorothiazide tablets — hydrochlorothiazide tablets may be administered orally, if necessary once daily, for up to 8 weeks

SUMMARY:
The initial 12 week portion of this 20 week study will examine the ability of a combination of olmesartan medoxomil and amlodipine to lower the blood pressure of patients with high blood pressure who have not had sufficient blood pressure reduction using one anti-hypertension drug (monotherapy). The final 8 weeks of this 20 week study will examine the ability of a combination of olmesartan medoxomil, amlodipine and hydrochlorothiazide to lower blood pressure in the same patient population. All three medications being tested have been approved by the FDA for the treatment of high blood pressure, but only amlodipine and olmesartan are currently approved for use in combination form.

ELIGIBILITY:
Inclusion Criteria:

* >= to 18 years of age
* Hypertension uncontrolled on current monotherapy
* Females:
* negative serum pregnancy test at screening
* post menopausal or have had a hysterectomy or tubal ligation or practicing approved methods of birth control

Exclusion Criteria:

* Pregnant females
* Uncontrolled hypertension with multiple drugs, except for hydrochlorothiazide/triamterene
* Diabetes requiring insulin
* Serious disorders that may limit the ability to evaluate the efficacy or safety of treatment
* History of myocardial infarction, bypass graft, angioplasty or heart failure within the past 6 months
* History of Class III or IV congestive heart failure
* History of stroke or transient ischemic attack within the last 1 year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 999 (Actual)
Dates: Start 2008-11; Primary Completion 2009-08 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (72):
- United States (72):
  - Birmingham, Alabama
  - Green Valley, Arizona
  - Mesa, Arizona
  - Sierra Vista, Arizona
  - Tempe, Arizona
  - Tucson, Arizona
  - Anaheim, California
  - Harbor City, California
  - National City, California
  - Tustin, California
  - Westlake Village, California
  - Colorado Springs, Colorado
  - Pueblo, Colorado
  - Milford, Connecticut
  - Boynton Beach, Florida
  - Brooksville, Florida
  - Clearwater, Florida
  - Deerfield Beach, Florida
  - DeLand, Florida
  - Fort Lauderdale, Florida
  - Kissimmee, Florida
  - Pembroke Pines, Florida
  - Sarasota, Florida
  - St. Petersburg, Florida
  - Tampa, Florida
  - Boise, Idaho
  - Addison, Illinois
  - Orland Park, Illinois
  - Wichita, Kansas
  - Lexington, Kentucky
  - Columbia, Maryland
  - Elkridge, Maryland
  - Oxon Hill, Maryland
  - Reisterstown, Maryland
  - Stevensville, Michigan
  - Omaha, Nebraska
  - Las Vegas, Nevada
  - Edison, New Jersey
  - Sewell, New Jersey
  - Albuquerque, New Mexico
  - Binghamton, New York
  - Cary, North Carolina
  - Charlotte, North Carolina
  - Harrisburg, North Carolina
  - Hickory, North Carolina
  - High Point, North Carolina
  - Raleigh, North Carolina
  - Wilmington, North Carolina
  - Winston-Salem, North Carolina
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Norman, Oklahoma
  - Oklahoma City, Oklahoma
  - Tulsa, Oklahoma
  - Eugene, Oregon
  - Portland, Oregon
  - Havertown, Pennsylvania
  - Jenkintown, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Greenville, South Carolina
  - Mt. Pleasant, South Carolina
  - New Tazewell, Tennessee
  - Amarillo, Texas
  - Austin, Texas
  - Carrollton, Texas
  - Corpus Christi, Texas
  - Dallas, Texas
  - Longview, Texas
  - West Jordan, Utah
  - Norfolk, Virginia
  - Walla Walla, Washington
  - Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/

REFERENCES:
- [Derived] Nesbitt SD, Shojaee A, Maa JF, Weir MR. Efficacy of an amlodipine/olmesartan treatment algorithm in patients with or without type 2 diabetes and hypertension (a secondary analysis of the BP-CRUSH study). J Hum Hypertens. 2013 Jul;27(7):445-52. doi: 10.1038/jhh.2012.65. Epub 2012 Dec 20. PMID 23254596
- [Derived] Hsueh WA, Shojaee A, Maa JF, Neutel JM. Efficacy of amlodipine/olmesartan medoxomil +/- HCTZ in obese patients uncontrolled on antihypertensive monotherapy. Curr Med Res Opin. 2012 Nov;28(11):1809-18. doi: 10.1185/03007995.2012.740632. Epub 2012 Oct 30. PMID 23072496

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred at approximately 140 outpatient medical clinics in the United States and South Africa from December 2008 through March 2009. 1406 uncontrolled hypertensive subjects were screened to place 999 subjects into active treatment.
Groups:
- Olmesartan Medoxomil/Amlodipine Tablets + Hydrochlorothiazide: Amlodipine and olmesartan medoxomil (Azor) oral tablets and hydrochlorothiazide oral tablets (if necessary) will be administered once a day for up to 20 weeks
Period: Overall Study
Arm/Group | Olmesartan Medoxomil/Amlodipine Tablets + Hydrochlorothiazide
Started | 999
Completed | 736
Not Completed | 263
Not completed — Adverse Event | 87
Not completed — Lost to Follow-up | 18
Not completed — Protocol Violation | 109
Not completed — Withdrawal by Subject | 40
Not completed — Did not take medication for >3 days | 1
Not completed — subject left area | 2
Not completed — non-compliance | 3
Not completed — Subject incarcerated | 1
Not completed — Subject required restricted medication | 1
Not completed — Lack of Efficacy | 1

BASELINE CHARACTERISTICS:
Arm/Group | Olmesartan Medoxomil/Amlodipine Tablets + Hydrochlorothiazide
Number analyzed (Participants) | 999
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 771
  >=65 years | 228
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 491
  Male | 508
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 6
  Asian | 129
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 234
  White | 630
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 732
  South Africa | 267
Hispanic or Latino [Number; unit: Participants]
  Hispanic or Latino | 105
  Non-Hispanic or Latino | 894
Type 2 Diabetes [Number; unit: Participants]
  Yes | 192
  No | 807
Weight [Mean (Standard Deviation); unit: kg] | 88.20 (21.466)
Body Mass Index [Mean (Standard Deviation); unit: Kg/m٨2] | 31.02 (6.370)
Metabolic syndrome [Number; unit: Participants] — Metabolic syndrome is defined as having at least 3 of the following parameters: waist circumference ≥40 inches (males) or ≥35 inches (females); triglycerides ≥150 mg/dL; high density lipoprotein cholesterol <40 mg/dL (males) or <50 mg/dL (females); blood pressure ≥130/85 mmHg; fasting glucose ≥100mg/dL; BMI ≥30kg/m2.
  Participants
    Yes | 462
    No | 537
Mean seated systolic blood pressure [Mean (Standard Deviation); unit: mm Hg] | 153.66 (9.178)
Mean seated diastolic blood pressure [Mean (Standard Deviation); unit: mm Hg] | 91.92 (8.616)
Pulse rate [Mean (Standard Deviation); unit: beats/minute] | 74.77 (11.621)
24-Hour mean systolic ambulatory blood pressure [Mean (Standard Deviation); unit: mm Hg] | 135.74 (11.698)
24-Hour mean diastolic ambulatory blood pressure [Mean (Standard Deviation); unit: mm Hg] | 81.09 (9.346)

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Patients Who Achieve Seated Systolic Blood Pressure Goal (<140 mm Hg for Non-diabetics and <130 mm Hg for Diabetics) From Baseline to 12 Weeks
Time Frame: baseline to 12 weeks
Population: The analysis population consists of those participants who have a baseline and at least 1 post-baseline measurement and who received at least one dose of study medication.
Measure: Number; unit: Percentage of participants
Arm/Group | Olmesartan Medoxomil/Amlodipine Tablets + Hydrochlorothiazide
Number analyzed (Participants) | 985
Percentage of participants | 75.8
Statistical Analysis 1: Comparison: Olmesartan Medoxomil/Amlodipine Tablets + Hydrochlorothiazide; Test type: Superiority or Other; Percentage = 75.8, 95% CI 2-sided [73.0 to 78.5]

2. Secondary Outcome: The Percentage of Subjects Achieving Seated Diastolic BP Goal (<90 mmHg for Non-diabetics or < 80 mmHg for Subjects With Diabetes) From Baseline to 12 Weeks
Time Frame: baseline to 12 weeks
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Olmesartan Medoxomil/Amlodipine Tablets + Hydrochlorothiazide
Number analyzed (Participants) | 985
Percentage of participants | 84.3
Statistical Analysis 1: Comparison: Olmesartan Medoxomil/Amlodipine Tablets + Hydrochlorothiazide; Test type: Superiority or Other; Percentage = 84.3, 95% CI 2-sided [81.8 to 86.5]

3. Secondary Outcome: The Percentage of Subjects Who Achieve BP Goal (<140/90 mmHg for Non-diabetics or <130/80 mmHg for Diabetics) From Baseline to 12 and 20 Weeks
Time Frame: Baseline to 12 and 20 weeks
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Olmesartan Medoxomil/Amlodipine Tablets + Hydrochlorothiazide
Number analyzed (Participants) | 985
Percentage of participants
  12 weeks | 71.3
  20 weeks | 84.8
Statistical Analysis 1: Comparison: Olmesartan Medoxomil/Amlodipine Tablets + Hydrochlorothiazide; 12 week analysis; Test type: Superiority or Other; Percentage = 71.3, 95% CI 2-sided [68.3 to 74.1]
Statistical Analysis 2: Comparison: Olmesartan Medoxomil/Amlodipine Tablets + Hydrochlorothiazide; 20 week analysis; Test type: Superiority or Other; Percentage = 84.8, 95% CI 2-sided [82.4 to 87.0]

4. Secondary Outcome: Change in Mean Seated Systolic Blood Pressure From Baseline to 4, 8, 12, 16, 20 Weeks
Time Frame: Baseline to 4, 8, 12, 16, 20 weeks
Population: The analysis population consists of those participants who have a baseline and at lease 1 post-baseline measurement and who received at least one dose of study medication. However, the number of participants included will vary because of missing data and the number of dropouts.
Measure: Mean (Standard Error); unit: mm Hg
Arm/Group | Olmesartan Medoxomil/Amlodipine Tablets + Hydrochlorothiazide
Number analyzed (Participants) | 975
mm Hg
  4 weeks, N=975 | -14.6 (0.42)
  8 weeks, N=929 | -16.6 (0.46)
  12 weeks, N=865 | -21.8 (0.46)
  16 weeks, N=797 | -26.0 (0.51)
  20 weeks, N=745 | -26.8 (0.53)
Statistical Analysis 1: Comparison: Olmesartan Medoxomil/Amlodipine Tablets + Hydrochlorothiazide; 4 week analysis; Test type: Superiority or Other; p < 0.0001, t-test, 1 sided; Median Difference (Net) = -14.6, 95% CI 2-sided [-15.4 to -13.8]
Statistical Analysis 2: Comparison: Olmesartan Medoxomil/Amlodipine Tablets + Hydrochlorothiazide; 8 week analysis; Test type: Superiority or Other; p < 0.0001, t-test, 1 sided; Mean Difference (Net) = -16.6, 95% CI 2-sided [-17.7 to -15.7]
Statistical Analysis 3: Comparison: Olmesartan Medoxomil/Amlodipine Tablets + Hydrochlorothiazide; 12 week analysis; Test type: Superiority or Other; p < 0.0001, t-test, 1 sided; Mean Difference (Net) = -21.8, 95% CI 2-sided [-22.7 to -20.9]
Statistical Analysis 4: Comparison: Olmesartan Medoxomil/Amlodipine Tablets + Hydrochlorothiazide; 16 week analysis; Test type: Superiority or Other; p < 0.0001, t-test, 1 sided; Mean Difference (Net) = -26.0, 95% CI 2-sided [-27.0 to -25.0]
Statistical Analysis 5: Comparison: Olmesartan Medoxomil/Amlodipine Tablets + Hydrochlorothiazide; 20 week analysis; Test type: Superiority or Other; p < 0.0001, t-test, 1 sided; Mean Difference (Net) = -26.8, 95% CI 2-sided [-27.8 to -25.7]

5. Secondary Outcome: Change in Mean Seated Diastolic Blood Pressure From Baseline to 4, 8, 12, 16, 20 Weeks
Time Frame: Baseline to 4, 8, 12, 16, 20 weeks
Population: The analysis population consists of those participants who have a baseline and at least 1 post-baseline measurement and who received at least one dose of study medication. However, the number of participants included will vary because of missing data and the number of dropouts.
Measure: Mean (Standard Error); unit: mm Hg
Arm/Group | Olmesartan Medoxomil/Amlodipine Tablets + Hydrochlorothiazide
Number analyzed (Participants) | 975
mm Hg
  4 weeks, N=975 | -8.1 (0.27)
  8 weeks, N=929 | -9.1 (0.29)
  12 weeks, N=865 | -11.9 (0.28)
  16 weeks, N=797 | -14.6 (0.31)
  20 weeks, N=745 | -14.5 (0.34)
Statistical Analysis 1: Comparison: Olmesartan Medoxomil/Amlodipine Tablets + Hydrochlorothiazide; 4 week analysis; Test type: Superiority or Other; p < 0.0001, t-test, 1 sided; Mean Difference (Net) = -8.1, 95% CI 2-sided [-8.6 to -7.6]
Statistical Analysis 2: Comparison: Olmesartan Medoxomil/Amlodipine Tablets + Hydrochlorothiazide; 8 week analysis; Test type: Superiority or Other; p < 0.0001, t-test, 1 sided; Mean Difference (Net) = -9.1, 95% CI 2-sided [-9.7 to -8.5]
Statistical Analysis 3: Comparison: Olmesartan Medoxomil/Amlodipine Tablets + Hydrochlorothiazide; 12 week analysis; Test type: Superiority or Other; p < 0.0001, t-test, 1 sided; Mean Difference (Net) = -11.9, 95% CI 2-sided [-12.5 to -11.4]
Statistical Analysis 4: Comparison: Olmesartan Medoxomil/Amlodipine Tablets + Hydrochlorothiazide; 16 week analysis; Test type: Superiority or Other; p < 0.0001, t-test, 1 sided; Mean Difference (Net) = -14.6, 95% CI 2-sided [-15.2 to -14.0]
Statistical Analysis 5: Comparison: Olmesartan Medoxomil/Amlodipine Tablets + Hydrochlorothiazide; 20 week analysis; Test type: Superiority or Other; p = 0.0001, t-test, 1 sided; Mean Difference (Net) = -14.5, 95% CI 2-sided [-15.1 to -13.8]

6. Secondary Outcome: Percentage of Patients Achieving Seated Diastolic Blood Pressure Goal From Baseline to 4, 8, 12, 16, 20 Weeks
Time Frame: Baseline to 4, 8, 12, 16, 20 weeks
Population: as for outcome 5
Measure: Number; unit: Percentage of participants
Arm/Group | Olmesartan Medoxomil/Amlodipine Tablets + Hydrochlorothiazide
Number analyzed (Participants) | 975
Percentage of participants
  4 weeks: <90 mm Hg, N=975 | 71.3
  4weeks: <85 mm Hg, N=975 | 55.2
  4 weeks: <80 mm Hg, N=975 | 34.2
  8 weeks: <90 mm Hg, N=929 | 75.1
  8 weeks: <85 mm Hg, N=929 | 57.1
  8 weeks: <80 mm Hg, N=929 | 40.2
  12 weeks: <90 mm Hg, N=865 | 84.3
  12 weeks: <85 mm Hg, N=865 | 68.7
  12 weeks: <80 mm Hg, N=865 | 49.5
  16 weeks: <90 mm Hg, N=797 | 90.2
  16 weeks: <85 mm Hg, N=797 | 76.9
  16 weeks: <80 mm Hg, N=797 | 59.6
  20 weeks: <90 mm Hg, N=745 | 89.7
  20 weeks: <85 mm Hg, N=745 | 79.5
  20 weeks: <80 mm Hg, N=745 | 62.0

7. Secondary Outcome: Percentage of Patients Achieving Seated Systolic Blood Pressure Goal From Baseline to 4, 8, 12, 16, 20 Weeks
Time Frame: Baseline to 4, 8, 12, 16, 20 weeks
Population: as for outcome 5
Measure: Number; unit: Percentage of Participants
Arm/Group | Olmesartan Medoxomil/Amlodipine Tablets + Hydrochlorothiazide
Number analyzed (Participants) | 975
Percentage of Participants
  4 weeks: <140 mm Hg, N=975 | 54.2
  4 weeks: <135 mm Hg, N=975 | 39.8
  4 weeks: <130 mm Hg, N=975 | 25.3
  4 weeks: <120 mm Hg, N=975 | 8.9
  8 weeks: <140 mm Hg, N=929 | 57.2
  8 weeks: <135 mm Hg, N=929 | 45.9
  8 weeks: <130 mm Hg, N=929 | 35.0
  8 weeks: <120 mm Hg, N=929 | 12.9
  12 weeks: <140 mm Hg, N=865 | 72.6
  12 weeks: <135 mm Hg, N=865 | 59.0
  12 weeks: <130 mm Hg, N=865 | 45.3
  12 weeks: <120 mm Hg, N=865 | 19.4
  16 weeks: <140 mm Hg, N=797 | 80.9
  16 weeks: <135 mm Hg, N=797 | 70.3
  16 weeks: <130 mm Hg, N=797 | 58.9
  16 weeks: <120 mm Hg, N=797 | 30.9
  20 weeks: <140 mm Hg, N=745 | 84.3
  20 weeks: <135 mm Hg, N=745 | 75.2
  20 weeks: <130 mm Hg, N=745 | 64.2
  20 weeks: <120 mm Hg, N=745 | 31.5

8. Secondary Outcome: Percentage of Patients Achieving Seated Blood Pressure Goal From Baseline to 4, 8, 12, 16, 20 Weeks
Time Frame: Baseline to 4, 8, 12, 16, 20 weeks
Population: as for outcome 5
Measure: Number; unit: Percentage of Participants
Arm/Group | Olmesartan Medoxomil/Amlodipine Tablets + Hydrochlorothiazide
Number analyzed (Participants) | 975
Percentage of Participants
  4 weeks: <140/90 mm Hg, N=975 | 49.1
  4 weeks: <135/80 mm Hg, N=975 | 23.0
  4 weeks: <130/80 mm Hg, N=975 | 17.3
  4 weeks: <120/80 mm Hg, N=975 | 7.8
  8 weeks: <140/90 mm Hg, N=929 | 52.4
  8 weeks: <135/80 mm Hg, N=929 | 29.8
  8 weeks: <130/80 mm Hg, N=929 | 24.8
  8 weeks: <120/80 mm Hg, N=929 | 11.2
  12 weeks: <140/90 mm Hg, N=865 | 68.1
  12 weeks: <135/80 mm Hg, N=865 | 40.0
  12 weeks: <130/80 mm Hg, N=865 | 34.3
  12 weeks: <120/80 mm Hg, N=865 | 17.6
  16 weeks: <140/90mm Hg, N=797 | 77.8
  16 weeks: <135/80mm Hg, N=797 | 51.3
  16 weeks: <130/80mm Hg, N=797 | 46.2
  16 weeks: <120/80mm Hg, N=797 | 28.7
  20 weeks: <140/90 mm Hg, N=745 | 81.3
  20 weeks: <135/80 mm Hg, N=745 | 55.6
  20 weeks: <130/80 mm Hg, N=745 | 50.1
  20 weeks: <120/80 mm Hg, N=745 | 28.2

9. Secondary Outcome: Percentage of Patients Achieving Seated Systolic Blood Pressure Reduction Ranges From Baseline to 4, 8, 12, 16, 20 Weeks
Time Frame: Baseline to 4, 8, 12, 16, 20 weeks
Population: as for outcome 5
Measure: Number; unit: Percentage of Participants
Arm/Group | Olmesartan Medoxomil/Amlodipine Tablets + Hydrochlorothiazide
Number analyzed (Participants) | 975
Percentage of Participants
  4 weeks: ≤ 15 mm Hg, N=975 | 51.4
  4 weeks: >15 and ≤ 30 mm Hg, N=975 | 36.6
  4 weeks: >30 and ≤ 45 mm Hg, N=975 | 10.5
  4 weeks: >45 mm Hg, N=975 | 1.5
  8 weeks: ≤ 15 mm Hg, N=929 | 45.8
  8 weeks: >15 and ≤ 30 mm Hg, N=929 | 37.7
  8 weeks: >30 and ≤ 45 mm Hg, N=929 | 14.3
  8 weeks: >45 mm Hg, N=929 | 2.3
  12 weeks: ≤ 15 mm Hg, N=865 | 30.5
  12 weeks: >15 and ≤ 30 mm Hg, N=865 | 43.1
  12 weeks: >30 and ≤ 45 mm Hg, N=865 | 22.4
  12 weeks: >45 mm Hg, N=865 | 3.9
  16 weeks: ≤ 15 mm Hg, N=797 | 23.2
  16 weeks: >15 and ≤ 30 mm Hg, N=797 | 35.9
  16 weeks: >30 and ≤ 45 mm Hg, N=797 | 32.0
  16 weeks: >45 mm Hg, N=797 | 8.9
  20 weeks: ≤ 15 mm Hg, N=745 | 20.4
  20 weeks: >15 and ≤ 30 mm Hg, N=745 | 36.2
  20 weeks: >30 and ≤ 45 mm Hg, N=745 | 34.0
  20 weeks: >45 mm Hg, N=745 | 9.4

10. Secondary Outcome: Percentage of Patients Achieving Seated Diastolic Blood Pressure Reduction Ranges From Baseline to 4, 8, 12, 16, 20 Weeks
Time Frame: Baseline to 4, 8, 12, 16, 20 weeks
Population: as for outcome 5
Measure: Number; unit: Percentage of Participants
Arm/Group | Olmesartan Medoxomil/Amlodipine Tablets + Hydrochlorothiazide
Number analyzed (Participants) | 975
Percentage of Participants
  4 weeks: ≤ 10 mm Hg, N=975 | 61.3
  4 weeks: >10 and ≤ 15 mm Hg, N=975 | 21.0
  4 weeks: >15 and ≤ 20 mm Hg, N=975 | 10.5
  4 weeks: >20 mm Hg, N=975 | 7.2
  8 weeks: ≤ 10 mm Hg, N=929 | 54.7
  8 weeks: >10 and ≤ 15 mm Hg, N=929 | 20.7
  8 weeks: >15 and ≤ 20 mm Hg, N=929 | 14.1
  8 weeks: >20 mm Hg, N=929 | 10.6
  12 weeks: ≤ 10 mm Hg, N=865 | 43.8
  12 weeks: >10 and ≤ 15 mm Hg, N=865 | 24.1
  12 weeks: >15 and ≤ 20 mm Hg, N=865 | 15.8
  12 weeks: >20 mm Hg, N=865 | 16.3
  16 weeks: ≤ 10 mm Hg, N=797 | 30.4
  16 weeks: >10 and ≤ 15 mm Hg, N=797 | 22.8
  16 weeks: >15 and ≤ 20 mm Hg, N=797 | 21.5
  16 weeks: >20 mm Hg, N=797 | 25.4
  20 weeks: ≤ 10 mm Hg, N=745 | 31.4
  20 weeks: >10 and ≤ 15 mm Hg, N=745 | 19.9
  20 weeks: >15 and ≤ 20 mm Hg, N=745 | 22.6
  20 weeks: >20 mm Hg, N=745 | 26.2

11. Secondary Outcome: Percentage of Participants Achieving the Mean Daytime Blood Pressure Goals, as Measured by Ambulatory Blood Pressure Monitor, From Baseline to 12 Weeks
Description: Once the Ambulatory Blood Pressure Monitor (ABPM) has been applied, the dose of medication was taken and the subject wore the ABPM for a period of 24 hours. Daytime is defined as 8AM - 4PM.
Time Frame: Baseline to 12 weeks
Population: Ambulatory blood pressure (ABPM) subset of participants who have both technically successful baseline and 12 week ABPM data.
Measure: Number; unit: Percentage of participants
Arm/Group | Olmesartan Medoxomil/Amlodipine Tablets + Hydrochlorothiazide
Number analyzed (Participants) | 229
Percentage of participants
  Daytime mean systolic blood pressure <140 mmHg | 88.2
  Daytime mean systolic blood pressure <135 mmHg | 79.9
  Daytime mean systolic blood pressure <130 mmHg | 66.4
  Daytime mean systolic blood pressure <120 mmHg | 28.8
  Daytime mean diastolic blood pressure <90 mmHg | 95.6
  Daytime mean diastolic blood pressure <85 mmHg | 83.0
  Daytime mean diastolic blood pressure <80 mmHg | 65.5
  Daytime mean blood pressure <140/90 mmHg | 86.9
  Daytime mean blood pressure <135/95 mmHg | 72.9
  Daytime mean blood pressure <135/80 mmHg | 61.1
  Daytime mean blood pressure <130/80 mmHg | 53.3
  Daytime mean blood pressure <125/75 mmHg | 31.9
  Daytime mean blood pressure <120/80 mmHg | 27.9
  Daytime mean blood pressure <120/70 mmHg | 13.1

12. Secondary Outcome: Percentage of Participants Achieving the Mean Daytime Blood Pressure Goals, as Measured by Ambulatory Blood Pressure Monitor, From Baseline to 20 Weeks
Description: as for outcome 11
Time Frame: Baseline to 20 weeks
Population: Ambulatory blood pressure (ABPM) subset of participants who have both technically successful baseline and 20 week ABPM data.
Measure: Number; unit: Percentage of participants
Arm/Group | Olmesartan Medoxomil/Amlodipine Tablets + Hydrochlorothiazide
Number analyzed (Participants) | 199
Percentage of participants
  Daytime mean systolic blood pressure <140 mmHg | 96.5
  Daytime mean systolic blood pressure <135 mmHg | 93.5
  Daytime mean systolic blood pressure <130 mmHg | 83.9
  Daytime mean systolic blood pressure <120 mmHg | 51.8
  Daytime mean diastolic blood pressure <90 mmHg | 98.5
  Daytime mean diastolic blood pressure <85 mmHg | 92.5
  Daytime mean diastolic blood pressure <80 mmHg | 83.9
  Daytime mean blood pressure <140/90 mmHg | 95.0
  Daytime mean blood pressure <135/95 mmHg | 88.4
  Daytime mean blood pressure <135/80 mmHg | 81.9
  Daytime mean blood pressure <130/80 mmHg | 77.4
  Daytime mean blood pressure <125/75 mmHg | 56.8
  Daytime mean blood pressure <120/80 mmHg | 51.3
  Daytime mean blood pressure <120/70 mmHg | 33.2

13. Secondary Outcome: Percentage of Participants Achieving the Mean Nighttime Blood Pressure Goals, as Measured by Ambulatory Blood Pressure Monitor, From Baseline to 12 Weeks
Description: Once the Ambulatory Blood Pressure Monitor (ABPM) has been applied, the dose of medication was taken and the subject wore the ABPM for a period of 24 hours. Nighttime is defined as 10p.m. - 6 a.m.
Time Frame: Baseline to 12 weeks
Population: as for outcome 11
Measure: Number; unit: Percentage of participants
Arm/Group | Olmesartan Medoxomil/Amlodipine Tablets + Hydrochlorothiazide
Number analyzed (Participants) | 229
Percentage of participants
  Nighttime mean systolic blood pressure <140 mmHg | 97.8
  Nighttime mean systolic blood pressure <135 mmHg | 94.3
  Nighttime mean systolic blood pressure <130 mmHg | 92.6
  Nighttime mean systolic blood pressure <120 mmHg | 74.7
  Nighttime mean diastolic blood pressure <90 mmHg | 99.6
  Nighttime mean diastolic blood pressure <85 mmHg | 98.3
  Nighttime mean diastolic blood pressure <80 mmHg | 94.8
  Nighttime mean blood pressure <140/90 mmHg | 97.4
  Nighttime mean blood pressure <135/95 mmHg | 93.4
  Nighttime mean blood pressure <135/80 mmHg | 90.8
  Nighttime mean blood pressure <130/80 mmHg | 89.1
  Nighttime mean blood pressure <125/75 mmHg | 77.7
  Nighttime mean blood pressure <120/80 mmHg | 74.2
  Nighttime mean blood pressure <120/70 mmHg | 62.0

14. Secondary Outcome: Percentage of Participants Achieving the Mean Nighttime Blood Pressure Goals, as Measured by Ambulatory Blood Pressure Monitor, From Baseline to 20 Weeks
Description: Once the Ambulatory Blood Pressure Monitor (ABPM) has been applied, the dose of medication was taken and the subject wore the ABPM for a period of 24 hours. Nighttime is defined as 10 p.m. - 6 a.m.
Time Frame: Baseline to 20 weeks
Population: as for outcome 12
Measure: Number; unit: Percentage of participants
Arm/Group | Olmesartan Medoxomil/Amlodipine Tablets + Hydrochlorothiazide
Number analyzed (Participants) | 199
Percentage of participants
  Nighttime mean systolic blood pressure <140 mmHg | 99.5
  Nighttime mean systolic blood pressure <135 mmHg | 99.5
  Nighttime mean systolic blood pressure <130 mmHg | 97.5
  Nighttime mean systolic blood pressure <120 mmHg | 86.4
  Nighttime mean diastolic blood pressure <90 mmHg | 99.5
  Nighttime mean diastolic blood pressure <85 mmHg | 98.5
  Nighttime mean diastolic blood pressure <80 mmHg | 96.0
  Nighttime mean blood pressure <140/90 mmHg | 99.0
  Nighttime mean blood pressure <135/95 mmHg | 98.5
  Nighttime mean blood pressure <135/80 mmHg | 96.0
  Nighttime mean blood pressure <130/80 mmHg | 95.0
  Nighttime mean blood pressure <125/75 mmHg | 88.9
  Nighttime mean blood pressure <120/80 mmHg | 85.9
  Nighttime mean blood pressure <120/70 mmHg | 78.9

15. Secondary Outcome: Percentage of Participants Achieving the Mean 24-hour Blood Pressure Goals, as Measured by Ambulatory Blood Pressure Monitor, From Baseline to 12 Weeks
Description: Once the Ambulatory Blood Pressure Monitor (ABPM) has been applied, the dose of medication was taken and the subject wore the ABPM for a period of 24 hours.
Time Frame: Baseline to 12 weeks
Population: as for outcome 11
Measure: Number; unit: Percentage of participants
Arm/Group | Olmesartan Medoxomil/Amlodipine Tablets + Hydrochlorothiazide
Number analyzed (Participants) | 229
Percentage of participants
  24-hour mean systolic blood pressure <140 mmHg | 95.6
  24-hour mean systolic blood pressure <135 mmHg | 90.4
  24-hour mean systolic blood pressure <130 mmHg | 79.9
  24-hour mean systolic blood pressure <120 mmHg | 47.2
  24-hour mean diastolic blood pressure <90 mmHg | 98.7
  24-hour mean diastolic blood pressure <85 mmHg | 96.1
  24-hour mean diastolic blood pressure <80 mmHg | 84.7
  24-hour mean blood pressure <140/90 mmHg | 94.3
  24-hour mean blood pressure <135/95 mmHg | 89.1
  24-hour mean blood pressure <135/80 mmHg | 80.3
  24-hour mean blood pressure <130/80 mmHg | 73.4
  24-hour mean blood pressure <125/75 mmHg | 52.4
  24-hour mean blood pressure <120/80 mmHg | 45.9
  24-hour mean blood pressure <120/70 mmHg | 27.5

16. Secondary Outcome: Percentage of Participants Achieving the Mean 24-hour Blood Pressure Goals, as Measured by Ambulatory Blood Pressure Monitor, From Baseline to 20 Weeks
Description: as for outcome 15
Time Frame: Baseline to 20 weeks
Population: as for outcome 12
Measure: Number; unit: Percentage of participants
Arm/Group | Olmesartan Medoxomil/Amlodipine Tablets + Hydrochlorothiazide
Number analyzed (Participants) | 199
Percentage of participants
  24-hour mean systolic blood pressure <140 mmHg | 99.5
  24-hour mean systolic blood pressure <135 mmHg | 97.5
  24-hour mean systolic blood pressure <130 mmHg | 94.5
  24-hour mean systolic blood pressure <120 mmHg | 70.4
  24-hour mean diastolic blood pressure <90 mmHg | 100.0
  24-hour mean diastolic blood pressure <85 mmHg | 97.5
  24-hour mean diastolic blood pressure <80 mmHg | 93.0
  24-hour mean blood pressure <140/90 mmHg | 99.5
  24-hour mean blood pressure <135/95 mmHg | 96.0
  24-hour mean blood pressure <135/80 mmHg | 92.5
  24-hour mean blood pressure <130/80 mmHg | 90.5
  24-hour mean blood pressure <125/75 mmHg | 75.4
  24-hour mean blood pressure <120/80 mmHg | 70.4
  24-hour mean blood pressure <120/70 mmHg | 55.3

17. Secondary Outcome: Change From Baseline to Week 12 in Ambulatory Systolic and Diastolic Blood Pressure Values
Description: Once the Ambulatory Blood Pressure Monitor (ABPM) has been applied, the dose of medication was taken and the subject wore the ABPM for a period of 24 hours. Daytime is defined as 8 a.m. to 4 p.m. Nighttime is defined as 10 p.m. to 6 a.m.
Time Frame: Baseline to 12 weeks
Population: as for outcome 11
Measure: Mean (Standard Error); unit: mm Hg
Arm/Group | Olmesartan Medoxomil/Amlodipine Tablets + Hydrochlorothiazide
Number analyzed (Participants) | 229
mm Hg
  24-hour mean systolic blood pressure | -14.8 (0.72)
  Mean daytime systolic blood pressure | -16.3 (0.77)
  Mean nighttime systolic blood pressure | -12.5 (0.84)
  Systolic blood pressure - last 2 hours of dose | -13.6 (1.04)
  Systolic blood pressure - last 4 hours of dose | -13.0 (0.90)
  Systolic blood pressure - last 6 hours of dose | -12.6 (0.85)
  24-hour mean diastolic blood pressure | -9.4 (0.46)
  Mean daytime diastolic blood pressure | -10.6 (0.51)
  Mean nighttime diastolic blood pressure | -7.6 (0.59)
  Diastolic blood pressure - last 2 hours of dose | -8.6 (0.70)
  Diastolic blood pressure - last 4 hours of dose | -8.0 (0.60)
  Diastolic blood pressure - last 6 hours of dose | -7.7 (0.57)
Statistical Analysis 1: Comparison: Olmesartan Medoxomil/Amlodipine Tablets + Hydrochlorothiazide; Mean 24-hour systolic blood pressure; Test type: Superiority or Other; p < 0.0001, t-test, 1 sided; Mean Difference (Net) = -14.8, 95% CI 2-sided [-16.2 to -13.4]
Statistical Analysis 2: Comparison: Olmesartan Medoxomil/Amlodipine Tablets + Hydrochlorothiazide; Mean daytime systolic blood pressure; Test type: Superiority or Other; p < 0.0001, t-test, 1 sided; Mean Difference (Net) = -16.3, 95% CI 2-sided [-17.8 to -14.8]
Statistical Analysis 3: Comparison: Olmesartan Medoxomil/Amlodipine Tablets + Hydrochlorothiazide; Mean nighttime systolic blood pressure; Test type: Superiority or Other; p < 0.0001, t-test, 1 sided; Mean Difference (Net) = -12.5, 95% CI 2-sided [-14.1 to -10.8]
Statistical Analysis 4: Comparison: Olmesartan Medoxomil/Amlodipine Tablets + Hydrochlorothiazide; systolic blood pressure during last 2 hours of dose; Test type: Superiority or Other; p < 0.0001, t-test, 1 sided; Mean Difference (Net) = -13.6, 95% CI 2-sided [-15.7 to -11.6]
Statistical Analysis 5: Comparison: Olmesartan Medoxomil/Amlodipine Tablets + Hydrochlorothiazide; systolic blood pressure during last 4 hours of dose; Test type: Superiority or Other; p < 0.0001, t-test, 1 sided; Mean Difference (Net) = -13.0, 95% CI 2-sided [-14.7 to -11.2]
Statistical Analysis 6: Comparison: Olmesartan Medoxomil/Amlodipine Tablets + Hydrochlorothiazide; systolic blood pressure during last 6 hours of dose; Test type: Superiority or Other; p < 0.0001, t-test, 1 sided; Mean Difference (Net) = -12.6, 95% CI 2-sided [-14.3 to -10.9]
Statistical Analysis 7: Comparison: Olmesartan Medoxomil/Amlodipine Tablets + Hydrochlorothiazide; Mean 24-hour diastolic blood pressure; Test type: Superiority or Other; p < 0.0001, t-test, 1 sided; Mean Difference (Net) = -9.4, 95% CI [-10.3 to -8.5]
Statistical Analysis 8: Comparison: Olmesartan Medoxomil/Amlodipine Tablets + Hydrochlorothiazide; Mean daytime diastolic blood pressure; Test type: Superiority or Other; p < 0.0001, t-test, 1 sided; Mean Difference (Net) = -10.6, 95% CI 2-sided [-11.7 to -9.6]
Statistical Analysis 9: Comparison: Olmesartan Medoxomil/Amlodipine Tablets + Hydrochlorothiazide; Mean nighttime diastolic blood pressure; Test type: Superiority or Other; p < 0.0001, t-test, 1 sided; Mean Difference (Net) = -7.6, 95% CI 2-sided [-8.8 to -6.4]
Statistical Analysis 10: Comparison: Olmesartan Medoxomil/Amlodipine Tablets + Hydrochlorothiazide; diastolic blood pressure during last 2 hours of dose; Test type: Superiority or Other; p < 0.0001, t-test, 1 sided; Mean Difference (Net) = -8.6, 95% CI [-10.0 to -7.2]
Statistical Analysis 11: Comparison: Olmesartan Medoxomil/Amlodipine Tablets + Hydrochlorothiazide; diastolic blood pressure during last 4 hours of dose; Test type: Superiority or Other; p < 0.0001, t-test, 1 sided; Mean Difference (Net) = -8.0, 95% CI 2-sided [-9.2 to -6.8]
Statistical Analysis 12: Comparison: Olmesartan Medoxomil/Amlodipine Tablets + Hydrochlorothiazide; diastolic blood pressure during last 6 hours of dose; Test type: Superiority or Other; p < 0.0001, t-test, 1 sided; Mean Difference (Net) = -7.7, 95% CI [-8.8 to -6.6]

18. Secondary Outcome: Change From Baseline to Week 20 in Ambulatory Systolic and Diastolic Blood Pressure Values
Description: as for outcome 17
Time Frame: Baseline to 20 weeks
Population: as for outcome 12
Measure: Mean (Standard Error); unit: mm Hg
Arm/Group | Olmesartan Medoxomil/Amlodipine Tablets + Hydrochlorothiazide
Number analyzed (Participants) | 199
mm Hg
  24-hour mean systolic blood pressure | -21.0 (0.84)
  Mean daytime systolic blood pressure | -23.2 (0.94)
  Mean nighttime systolic blood pressure | -17.5 (0.94)
  Systolic blood pressure - last 2 hours of dose | -19.6 (1.10)
  Systolic blood pressure - last 4 hours of dose | -18.2 (1.00)
  Systolic blood pressure - last 6 hours of dose | -17.9 (0.95)
  24-hour mean diastolic blood pressure | -13.3 (0.55)
  Mean daytime diastolic blood pressure | -15.0 (0.62)
  Mean nighttime diastolic blood pressure | -11.1 (0.69)
  Diastolic blood pressure - last 2 hours of dose | -12.3 (0.77)
  Diastolic blood pressure - last 4 hours of dose | -11.6 (0.69)
  Diastolic blood pressure - last 6 hours of dose | -11.3 (0.66)
Statistical Analysis 1: Comparison: Olmesartan Medoxomil/Amlodipine Tablets + Hydrochlorothiazide; 24-hour mean systolic blood pressure; Test type: Superiority or Other; p < 0.0001, t-test, 1 sided; Mean Difference (Net) = -21.0, 95% CI 2-sided [-22.6 to -19.3]
Statistical Analysis 2: Comparison: Olmesartan Medoxomil/Amlodipine Tablets + Hydrochlorothiazide; Mean daytime systolic blood pressure; Test type: Superiority or Other; p < 0.0001, t-test, 1 sided; Mean Difference (Net) = -23.2, 95% CI 2-sided [-25.1 to -21.4]
Statistical Analysis 3: Comparison: Olmesartan Medoxomil/Amlodipine Tablets + Hydrochlorothiazide; Mean nighttime systolic blood pressure; Test type: Superiority or Other; p < 0.0001, t-test, 1 sided; Mean Difference (Net) = -17.5, 95% CI 2-sided [-19.4 to -15.6]
Statistical Analysis 4: Comparison: Olmesartan Medoxomil/Amlodipine Tablets + Hydrochlorothiazide; Systolic blood pressure - last 2 hours of dose; Test type: Superiority or Other; p < 0.0001, t-test, 1 sided; Mean Difference (Net) = -19.6, 95% CI 2-sided [-21.7 to -17.4]
Statistical Analysis 5: Comparison: Olmesartan Medoxomil/Amlodipine Tablets + Hydrochlorothiazide; Systolic blood pressure - last 4 hours of dose; Test type: Superiority or Other; p < 0.0001, t-test, 1 sided; Mean Difference (Net) = -18.2, 95% CI 2-sided [-20.2 to -16.3]
Statistical Analysis 6: Comparison: Olmesartan Medoxomil/Amlodipine Tablets + Hydrochlorothiazide; Systolic blood pressure - last 6 hours of dose; Test type: Superiority or Other; p < 0.0001, t-test, 1 sided; Mean Difference (Net) = -17.9, 95% CI 2-sided [-19.7 to -16.0]
Statistical Analysis 7: Comparison: Olmesartan Medoxomil/Amlodipine Tablets + Hydrochlorothiazide; 24-hour mean diastolic blood pressure; Test type: Superiority or Other; p < 0.0001, t-test, 1 sided; Mean Difference (Net) = -13.3, 95% CI 2-sided [-14.4 to -12.2]
Statistical Analysis 8: Comparison: Olmesartan Medoxomil/Amlodipine Tablets + Hydrochlorothiazide; Mean daytime diastolic blood pressure; Test type: Superiority or Other; p < 0.0001, t-test, 1 sided; Mean Difference (Net) = -15.0, 95% CI 2-sided [-16.2 to -13.8]
Statistical Analysis 9: Comparison: Olmesartan Medoxomil/Amlodipine Tablets + Hydrochlorothiazide; Mean nighttime diastolic blood pressure; Test type: Superiority or Other; p < 0.0001, t-test, 1 sided; Mean Difference (Net) = -11.1, 95% CI 2-sided [-12.4 to -9.8]
Statistical Analysis 10: Comparison: Olmesartan Medoxomil/Amlodipine Tablets + Hydrochlorothiazide; Diastolic blood pressure - last 2 hours of dose; Test type: Superiority or Other; p < 0.0001, t-test, 1 sided; Mean Difference (Net) = -12.3, 95% CI 2-sided [-13.8 to -10.8]
Statistical Analysis 11: Comparison: Olmesartan Medoxomil/Amlodipine Tablets + Hydrochlorothiazide; Diastolic blood pressure - last 4 hours of dose; Test type: Superiority or Other; p < 0.0001, t-test, 1 sided; Mean Difference (Net) = -11.6, 95% CI 2-sided [-12.9 to -10.2]
Statistical Analysis 12: Comparison: Olmesartan Medoxomil/Amlodipine Tablets + Hydrochlorothiazide; Diastolic blood pressure - last 6 hours of dose; Test type: Superiority or Other; p < 0.0001, t-test, 1 sided; Mean Difference (Net) = -11.3, 95% CI 2-sided [-12.6 to -10.0]

19. Secondary Outcome: Percentage of African American/Black Patients Achieving Seated Systolic Blood Pressure Goal From Baseline to 4, 8, 12, 16, 20 Weeks
Time Frame: Baseline to 4, 8, 12, 16, 20 weeks
Population: The analysis population consists of those African American/Black participants who have a baseline and at least 1 post-baseline measurement and who received at least one dose of study medication. However, the number of participants included will vary because of missing data and the number of dropouts.
Measure: Number; unit: Percentage of Participants
Arm/Group | Olmesartan Medoxomil/Amlodipine Tablets + Hydrochlorothiazide
Number analyzed (Participants) | 230
Percentage of Participants
  4 weeks: <140 mm Hg, N=230 | 51.7
  4 weeks: <135 mm Hg, N=230 | 34.4
  4 weeks: <130 mm Hg, N=230 | 19.6
  4 weeks: <120 mm Hg, N=230 | 5.7
  8 weeks: <140 mm Hg, N=231 | 62.3
  8 weeks: <135 mm Hg, N=231 | 44.6
  8 weeks: <130 mm Hg, N=231 | 33.8
  8 weeks: <120 mm Hg, N=231 | 13.0
  12 weeks: <140 mm Hg, N=232 | 76.3
  12 weeks: <135 mm Hg, N=232 | 59.1
  12 weeks: <130 mm Hg, N=232 | 47.0
  12 weeks: <120 mm Hg, N=232 | 19.8
  16 weeks: <140 mm Hg, N=232 | 84.9
  16 weeks: <135 mm Hg, N=232 | 71.1
  16 weeks: <130 mm Hg, N=232 | 61.2
  16 weeks: <120 mm Hg, N=232 | 34.1
  20 weeks: <140 mm Hg, N=232 | 91.0
  20 weeks: <135 mm Hg, N=232 | 80.6
  20 weeks: <130 mm Hg, N=232 | 71.1
  20 weeks: <120 mm Hg, N=232 | 44.4

20. Secondary Outcome: Percentage of African American/Black Patients Achieving Seated Diastolic Blood Pressure Goal From Baseline to 4, 8, 12, 16, 20 Weeks
Time Frame: Baseline to 4, 8, 12, 16, 20 weeks
Population: as for outcome 19
Measure: Number; unit: Percentage of Participants
Arm/Group | Olmesartan Medoxomil/Amlodipine Tablets + Hydrochlorothiazide
Number analyzed (Participants) | 230
Percentage of Participants
  4 weeks: <90 mm Hg, N=230 | 60.9
  4 weeks: <85 mm Hg, N=230 | 42.2
  4 weeks: <80 mm Hg, N=230 | 19.6
  8 weeks: <90 mm Hg, N=231 | 71.9
  8 weeks: <85 mm Hg, N=231 | 53.7
  8 weeks: <80 mm Hg, N=231 | 30.3
  12 weeks: <90 mm Hg, N=232 | 82.3
  12 weeks: <85 mm Hg, N=232 | 66.0
  12 weeks: <80 mm Hg, N=232 | 45.3
  16 weeks: <90 mm Hg, N=232 | 92.2
  16 weeks: <85 mm Hg, N=232 | 76.3
  16 weeks: <80 mm Hg, N=232 | 55.2
  20 weeks: <90 mm Hg, N=232 | 94.8
  20 weeks: <85 mm Hg, N=232 | 80.6
  20 weeks: <80 mm Hg, N=232 | 61.2

21. Secondary Outcome: Percentage of African American/Black Patients Achieving Seated Blood Pressure Goal From Baseline to 4, 8, 12, 16, 20 Weeks
Time Frame: Baseline to 4, 8, 12, 16, 20 weeks
Population: as for outcome 19
Measure: Number; unit: Percentage of Participants
Arm/Group | Olmesartan Medoxomil/Amlodipine Tablets + Hydrochlorothiazide
Number analyzed (Participants) | 230
Percentage of Participants
  4 weeks: <140/90 mm Hg, N=230 | 45.7
  4 weeks: <135/80 mm Hg, N=230 | 14.8
  4 weeks: <130/80 mm Hg, N=230 | 10.4
  4 weeks: <120/80 mm Hg, N=230 | 3.9
  8 weeks: <140/90 mm Hg, N=231 | 55.0
  8 weeks: <135/80 mm Hg, N=231 | 23.8
  8 weeks: <130/80 mm Hg, N=232 | 20.8
  8 weeks: <120/80 mm Hg, N=232 | 10.4
  12 weeks: <140/90mm Hg, N=232 | 68.5
  12 weeks: <135/80 mm Hg, N=232 | 38.4
  12 weeks: <130/80 mm Hg, N=232 | 35.8
  12 weeks: <120/80 mm Hg, N=232 | 16.4
  16 weeks: <140/90 mm Hg, N=232 | 80.6
  16 weeks: <135/80 mm Hg, N=232 | 49.1
  16 weeks: <130/80 mm Hg, N=232 | 47.4
  16 weeks: <120/80 mm Hg, N=232 | 30.6
  20 weeks: <140/90 mm Hg, N=232 | 86.6
  20 weeks: <135/80 mm Hg, N=232 | 57.8
  20 weeks: <130/80 mm Hg, N=232 | 55.2
  20 weeks: <120/80 mm Hg, N=232 | 39.7

22. Secondary Outcome: Percentage of African American/Black Patients Achieving Seated Systolic Blood Pressure Reduction Ranges From Baseline to 4, 8, 12, 16, 20 Weeks
Time Frame: Baseline to 4, 8, 12, 16, 20 weeks
Population: as for outcome 5
Measure: Number; unit: Percentage of Participants
Arm/Group | Olmesartan Medoxomil/Amlodipine Tablets + Hydrochlorothiazide
Number analyzed (Participants) | 230
Percentage of Participants
  4 weeks: ≤ 15 mm Hg, N=230 | 60.0
  4 weeks: >15 and ≤ 30 mm Hg, N=230 | 32.2
  4 weeks: >30 and ≤ 45 mm Hg, N=230 | 7.4
  4 weeks: >45 mm Hg, N=230 | 0.4
  8 weeks: ≤ 15 mm Hg, N=220 | 53.6
  8 weeks: >15 and ≤ 30 mm Hg, N=220 | 38.2
  8 weeks: >30 and ≤ 45 mm Hg, N=220 | 7.3
  8 weeks: >45 mm Hg, N=220 | 0.9
  12 weeks: ≤ 15 mm Hg, N=208 | 38.9
  12 weeks: >15 and ≤ 30 mm Hg, N=208 | 41.8
  12 weeks: >30 and ≤ 45 mm Hg, N=208 | 16.4
  12 weeks: >45 mm Hg, N=208 | 2.9
  16 weeks: ≤ 15 mm Hg, N=199 | 30.7
  16 weeks: >15 and ≤ 30 mm Hg, N=199 | 37.2
  16 weeks: >30 and ≤ 45 mm Hg, N=199 | 25.1
  16 weeks: >45 mm Hg, N=199 | 7.0
  20 weeks: ≤ 15 mm Hg, N=189 | 24.3
  20 weeks: >15 and ≤ 30 mm Hg, N=189 | 37.6
  20 weeks: >30 and ≤ 45 mm Hg, N=189 | 29.6
  20 weeks: >45 mm Hg, N=189 | 8.5

23. Secondary Outcome: Percentage of African American/Black Patients Achieving Seated Diastolic Blood Pressure Reduction Ranges From Baseline to 4, 8, 12, 16, 20 Weeks
Time Frame: Baseline to 4, 8, 12, 16, 20 weeks
Population: as for outcome 5
Measure: Number; unit: Percentage of Participants
Arm/Group | Olmesartan Medoxomil/Amlodipine Tablets + Hydrochlorothiazide
Number analyzed (Participants) | 230
Percentage of Participants
  4 weeks: ≤ 10 mm Hg, N=230 | 70.0
  4 weeks: >10 and ≤ 15 mm Hg, N=230 | 17.8
  4 weeks: >15 and ≤ 20 mm Hg, N=230 | 7.9
  4 weeks: >20 mm Hg, N=230 | 4.4
  8 weeks: ≤ 10 mm Hg, N=220 | 66.8
  8 weeks: >10 and ≤ 15 mm Hg, N=220 | 15.0
  8 weeks: >15 and ≤ 20 mm Hg, N=220 | 10.9
  8 weeks: >20 mm Hg, N=220 | 7.3
  12 weeks: ≤ 10 mm Hg, N=208 | 54.8
  12 weeks: >10 and ≤15 mm Hg, N=208 | 21.2
  12 weeks: >15 and ≤ 20 mm Hg, N=208 | 12.0
  12 weeks: >20 mm Hg, N=208 | 12.0
  16 weeks: ≤ 10 mm Hg, N=199 | 38.7
  16 weeks: >10 and ≤ 15 mm Hg, N=199 | 19.6
  16 weeks: >15 and ≤ 20 mm Hg, N=199 | 23.1
  16 weeks: >20 mm Hg, N=199 | 18.6
  20 weeks: ≤ 10 mm Hg, N=189 | 36.0
  20 weeks: >10 and ≤ 15 mm Hg, N=189 | 19.6
  20 weeks: >15 and ≤ 20 mm Hg, N=189 | 20.6
  20 weeks: >20 mm Hg, N=189 | 23.8

24. Secondary Outcome: Percentage of Asian Patients Achieving Seated Systolic Blood Pressure Goal From Baseline to 4, 8, 12, 16, 20 Weeks
Time Frame: Baseline to 4, 8, 12, 16, 20 weeks
Population: The analysis population consists of those Asian participants who have a baseline and at least 1 post-baseline measurement and who received at least one dose of study medication. However, the number of participants included may vary because of missing data and the number of dropouts.
Measure: Number; unit: Percentage of Participants
Arm/Group | Olmesartan Medoxomil/Amlodipine Tablets + Hydrochlorothiazide
Number analyzed (Participants) | 128
Percentage of Participants
  4 weeks: <140 mm Hg, N=128 | 64.8
  4 weeks: <135 mm Hg, N=128 | 51.6
  4 weeks: <130 mm Hg, N=128 | 35.2
  4 weeks: <120 mm Hg, N=128 | 11.7
  8 weeks: <140 mm Hg, N=128 | 76.6
  8 weeks: <135 mm Hg, N=128 | 67.2
  8 weeks: <130 mm Hg, N=128 | 51.6
  8 weeks: <120 mm Hg, N=128 | 25.0
  12 weeks: <140 mm Hg, N=128 | 89.1
  12 weeks: <135 mm Hg, N=128 | 78.9
  12 weeks: <130 mm Hg, N=128 | 66.4
  12 weeks: <120 mm Hg, N=128 | 38.3
  16 weeks: <140 mm Hg, N=128 | 95.3
  16 weeks: <135 mm Hg, N=128 | 89.8
  16 weeks: <130 mm Hg, N=128 | 81.3
  16 weeks: <120 mm Hg, N=128 | 47.7
  20 weeks: <140 mm Hg, N=128 | 97.7
  20 weeks: <135 mm Hg, N=128 | 93.0
  20 weeks: <130 mm Hg, N=128 | 85.9
  20 weeks: <120 mm Hg, N=128 | 51.6

25. Secondary Outcome: Percentage of Asain Patients Achieving Seated Diastolic Blood Pressure Goal From Baseline to 4, 8, 12, 16, 20 Weeks
Time Frame: Baseline to 4, 8, 12, 16, 20 weeks
Population: The analysis population consists of those Asian participants who have a baseline and at least 1 post-baseline measurement and who received at least one dose of study medication. However, the number of participants included will vary because of missing data and the number of dropouts.
Measure: Number; unit: Percentage of Participants
Arm/Group | Olmesartan Medoxomil/Amlodipine Tablets + Hydrochlorothiazide
Number analyzed (Participants) | 128
Percentage of Participants
  4 weeks: <90 mm Hg, N=128 | 83.6
  4 weeks: <85 mm Hg, N=128 | 69.5
  4 weeks: <80 mm Hg, N=128 | 45.3
  8 weeks: <90 mm Hg, N=128 | 89.1
  8 weeks: <85 mm Hg, N=128 | 79.7
  8 weeks: <80 mm Hg, N=128 | 60.2
  12 weeks: <90 mm Hg, N=128 | 95.3
  12 weeks: <85 mm Hg, N=128 | 87.5
  12 weeks: <80 mm Hg, N=128 | 71.1
  16 weeks: <90 mm Hg, N=128 | 96.9
  16 weeks: <85 mm Hg, N=128 | 93.0
  16 weeks: <80 mm Hg, N=128 | 82.0
  20 weeks: <90 mm Hg, N=128 | 96.9
  20 weeks: <85 mm Hg, N=128 | 93.0
  20 weeks: <80 mm Hg, N=128 | 85.2

26. Secondary Outcome: Percentage of Asian Patients Achieving Seated Systolic Blood Pressure Reduction Ranges From Baseline to 4, 8, 12, 16, 20 Weeks
Time Frame: Baseline to 4, 8, 12, 16, 20 weeks
Population: as for outcome 25
Measure: Number; unit: Percentage of Participants
Arm/Group | Olmesartan Medoxomil/Amlodipine Tablets + Hydrochlorothiazide
Number analyzed (Participants) | 126
Percentage of Participants
  4 weeks: ≤ 15 mm Hg, N=126 | 43.7
  4 weeks: >15 and ≤ 30 mm Hg, N=126 | 38.1
  4 weeks: >30 and ≤ 45 mm Hg, N=126 | 15.9
  4 weeks: >45 mm Hg, N=126 | 2.4
  8 weeks: ≤ 15 mm Hg, N=123 | 40.7
  8 weeks: >15 and ≤ 30 mm Hg, N=123 | 35.8
  8 weeks: >30 and ≤ 45 mm Hg, N=123 | 22.0
  8 weeks: >45 mm Hg, N=123 | 1.6
  12 weeks: ≤ 15 mm Hg, N=120 | 28.3
  12 weeks: >15 and ≤ 30 mm Hg, N=120 | 39.2
  12 weeks: >30 and ≤ 45 mm Hg, N=120 | 27.5
  12 weeks: >45 mm Hg, N=120 | 5.0
  16 weeks: ≤ 15 mm Hg, N=112 | 20.5
  16 weeks: >15 and ≤ 30 mm Hg, N=112 | 36.6
  16 weeks: >30 and ≤ 45 mm Hg, N=112 | 31.3
  16 weeks: >45 mm Hg, N=112 | 11.6
  20 weeks: ≤ 15 mm Hg, N=105 | 29.5
  20 weeks: >15 and ≤ 30 mm Hg, N=105 | 28.6
  20 weeks: >30 and ≤ 45 mm Hg, N=105 | 33.3
  20 weeks: >45 mm Hg, N=105 | 8.6

27. Secondary Outcome: Percentage of Asian Patients Achieving Seated Diastolic Blood Pressure Reduction Ranges From Baseline to 4, 8, 12, 16, 20 Weeks
Time Frame: Baseline to 4, 8, 12, 16, 20 weeks
Population: as for outcome 25
Measure: Number; unit: Percentage of Participants
Arm/Group | Olmesartan Medoxomil/Amlodipine Tablets + Hydrochlorothiazide
Number analyzed (Participants) | 126
Percentage of Participants
  4 weeks: ≤ 10 mm Hg, N=126 | 47.6
  4 weeks: >10 and ≤ 15 mm Hg, N=126 | 26.2
  4 weeks: >15 and ≤ 20 mm Hg, N=126 | 13.5
  4 weeks: >20 mm Hg, N=126 | 12.7
  8 weeks: ≤ 10 mm Hg, N=123 | 38.2
  8 weeks: >10 and ≤ 15 mm Hg, N=123 | 24.4
  8 weeks: >15 and ≤ 20 mm Hg, N=123 | 22.0
  8 weeks: >20 mm Hg, N=123 | 15.5
  12 weeks: ≤ 10 mm Hg, N=120 | 33.3
  12 weeks: >10 and ≤15 mm Hg, N=120 | 25.8
  12 weeks: >15 and ≤ 20 mm Hg, N=120 | 19.2
  12 weeks: >20 mm Hg, N=120 | 21.7
  16 weeks: ≤ 10 mm Hg, N=112 | 27.7
  16 weeks: >10 and ≤ 15 mm Hg, N=112 | 17.0
  16 weeks: >15 and ≤ 20 mm Hg, N=112 | 20.5
  16 weeks: >20 mm Hg, N=112 | 34.8
  20 weeks: ≤ 10 mm Hg, N=105 | 36.2
  20 weeks: >10 and ≤ 15 mm Hg, N=105 | 16.2
  20 weeks: >15 and ≤ 20 mm Hg, N=105 | 18.1
  20 weeks: >20 mm Hg, N=105 | 29.5

28. Secondary Outcome: Percentage of Hispanic Patients Achieving Seated Systolic Blood Pressure Goal From Baseline to 4, 8, 12, 16, 20 Weeks
Time Frame: Baseline to 4, 8, 12, 16, 20 weeks
Population: The analysis population consists of those Hispanic participants who have a baseline and at least 1 post-baseline measurement and who received at least one dose of study medication. However, the number of participants included may vary because of missing data and the number of dropouts.
Measure: Number; unit: Percentage of Participants
Arm/Group | Olmesartan Medoxomil/Amlodipine Tablets + Hydrochlorothiazide
Number analyzed (Participants) | 98
Percentage of Participants
  4 weeks: <140 mm Hg, N=98 | 55.1
  4 weeks: <135 mm Hg, N=98 | 39.8
  4 weeks: <130 mm Hg, N=98 | 31.6
  4 weeks: <120 mm Hg, N=98 | 10.2
  8 weeks: <140 mm Hg, N=100 | 64.0
  8 weeks: <135 mm Hg, N=100 | 51.0
  8 weeks: <130 mm Hg, N=100 | 41.0
  8 weeks: <120 mm Hg, N=100 | 15.0
  12 weeks: <140 mm Hg, N=100 | 77.0
  12 weeks: <135 mm Hg, N=100 | 67.0
  12 weeks: <130 mm Hg, N=100 | 54.0
  12 weeks: <120 mm Hg, N=100 | 30.0
  16 weeks: <140 mm Hg, N=100 | 84.0
  16 weeks: <135 mm Hg, N=100 | 77.0
  16 weeks: <130 mm Hg, N=100 | 66.0
  16 weeks: <120 mm Hg, N=100 | 37.0
  20 weeks: <140 mm Hg, N=100 | 88.0
  20 weeks: <135 mm Hg, N=100 | 83.0
  20 weeks: <130 mm Hg, N=100 | 72.0
  20 weeks: <120 mm Hg, N=100 | 41.0

29. Secondary Outcome: Percentage of Hispanic Patients Achieving Seated Diastolic Blood Pressure Goal From Baseline to 4, 8, 12, 16, 20 Weeks
Time Frame: Baseline to 4, 8, 12, 16, 20 weeks
Population: The analysis population consists of those Hispanic participants who have a baseline and at least 1 post-baseline measurement and who received at least one dose of study medication. However, the number of participants included will vary because of missing data and the number of dropouts.
Measure: Number; unit: Percentage of Participants
Arm/Group | Olmesartan Medoxomil/Amlodipine Tablets + Hydrochlorothiazide
Number analyzed (Participants) | 98
Percentage of Participants
  4 weeks: <90 mm Hg, N=98 | 66.3
  4 weeks: <85 mm Hg, N=98 | 53.1
  4 weeks: <80 mm Hg, N=98 | 34.7
  8 weeks: <90 mm Hg, N=100 | 85.0
  8 weeks: <85 mm Hg, N=100 | 70.0
  8 weeks: <80 mm Hg, N=100 | 48.0
  12 weeks: <90 mm Hg, N=100 | 92.0
  12 weeks: <85 mm Hg, N=100 | 78.0
  12 weeks: <80 mm Hg, N=100 | 62.0
  16 weeks: <90 mm Hg, N=100 | 96.0
  16 weeks: <85 mm Hg, N=100 | 90.0
  16 weeks: <80 mm Hg, N=100 | 75.0
  20 weeks: <90 mm Hg, N=100 | 96.0
  20 weeks: <85 mm Hg, N=100 | 90.0
  20 weeks: <80 mm Hg, N=100 | 75.0

30. Secondary Outcome: Percentage of Hispanic Patients Achieving Seated Systolic Blood Pressure Reduction Ranges From Baseline to 4, 8, 12, 16, 20 Weeks
Time Frame: Baseline to 4, 8, 12, 16, 20 weeks
Population: as for outcome 29
Measure: Number; unit: Percentage of Participants
Arm/Group | Olmesartan Medoxomil/Amlodipine Tablets + Hydrochlorothiazide
Number analyzed (Participants) | 98
Percentage of Participants
  4 weeks: ≤ 15 mm Hg, N=98 | 50.0
  4 weeks: >15 and ≤ 30 mm Hg, N=98 | 37.8
  4 weeks: >30 and ≤ 45 mm Hg, N=98 | 7.1
  4 weeks: >45 mm Hg, N=98 | 5.1
  8 weeks: ≤ 15 mm Hg, N=91 | 42.9
  8 weeks: >15 and ≤ 30 mm Hg, N=91 | 44.0
  8 weeks: >30 and ≤ 45 mm Hg, N=91 | 9.9
  8 weeks: >45 mm Hg, N=91 | 3.3
  12 weeks: ≤ 15 mm Hg, N=83 | 31.3
  12 weeks: >15 and ≤ 30 mm Hg, N=83 | 36.1
  12 weeks: >30 and ≤ 45 mm Hg, N=83 | 25.3
  12 weeks: >45 mm Hg, N=83 | 7.2
  16 weeks: ≤ 15 mm Hg, N=75 | 22.7
  16 weeks: >15 and ≤ 30 mm Hg, N=75 | 36.0
  16 weeks: >30 and ≤ 45 mm Hg, N=75 | 34.7
  16 weeks: >45 mm Hg, N=75 | 6.7
  20 weeks: ≤ 15 mm Hg, N=71 | 23.9
  20 weeks: >15 and ≤ 30 mm Hg, N=71 | 33.8
  20 weeks: >30 and ≤ 45 mm Hg, N=71 | 33.8
  20 weeks: >45 mm Hg, N=71 | 8.5

31. Secondary Outcome: Percentage of Hispanic Patients Achieving Seated Diastolic Blood Pressure Reduction Ranges From Baseline to 4, 8, 12, 16, 20 Weeks
Time Frame: Baseline to 4, 8, 12, 16, 20 weeks
Population: as for outcome 29
Measure: Number; unit: Percentage of Participants
Arm/Group | Olmesartan Medoxomil/Amlodipine Tablets + Hydrochlorothiazide
Number analyzed (Participants) | 98
Percentage of Participants
  4 weeks: ≤ 10 mm Hg, N=98 | 65.3
  4 weeks: >10 and ≤ 15 mm Hg, N=98 | 16.3
  4 weeks: >15 and ≤ 20 mm Hg, N=98 | 8.2
  4 weeks: >20 mm Hg, N=98 | 10.2
  8 weeks: ≤ 10 mm Hg, N=91 | 52.8
  8 weeks: >10 and ≤ 15 mm Hg, N=91 | 18.7
  8 weeks: >15 and ≤ 20 mm Hg, N=91 | 14.3
  8 weeks: >20 mm Hg, N=91 | 14.3
  12 weeks: ≤ 10 mm Hg, N=83 | 41.0
  12 weeks: >10 and ≤15 mm Hg, N=83 | 20.5
  12 weeks: >15 and ≤ 20 mm Hg, N=83 | 14.5
  12 weeks: >20 mm Hg, N=83 | 24.1
  16 weeks: ≤ 10 mm Hg, N=75 | 30.7
  16 weeks: >10 and ≤ 15 mm Hg, N=75 | 25.3
  16 weeks: >15 and ≤ 20 mm Hg, N=75 | 16.0
  16 weeks: >20 mm Hg, N=75 | 28.0
  20 weeks: ≤ 10 mm Hg, N=71 | 31.0
  20 weeks: >10 and ≤ 15 mm Hg, N=71 | 12.7
  20 weeks: >15 and ≤ 20 mm Hg, N=71 | 26.8
  20 weeks: >20 mm Hg, N=71 | 29.6

32. Secondary Outcome: Percentage of Elderly Patients Achieving Seated Systolic Blood Pressure Goal From Baseline to 4, 8, 12, 16, 20 Weeks
Time Frame: Baseline to 4, 8, 12, 16, 20 weeks
Population: The analysis population consists of those elderly participants who have a baseline and at least 1 post-baseline measurement and who received at least one dose of study medication. However, the number of participants included may vary because of missing data and the number of dropouts. Elderly is defined as greater than or = to 65 years of age.
Measure: Number; unit: Percentage of Participants
Arm/Group | Olmesartan Medoxomil/Amlodipine Tablets + Hydrochlorothiazide
Number analyzed (Participants) | 227
Percentage of Participants
  4 weeks: <140 mm Hg, N=227 | 52.0
  4 weeks: <135 mm Hg, N=227 | 37.9
  4 weeks: <130 mm Hg, N=227 | 23.4
  4 weeks: <120 mm Hg, N=227 | 9.7
  8 weeks: <140 mm Hg, N=227 | 67.0
  8 weeks: <135 mm Hg, N=227 | 57.7
  8 weeks: <130 mm Hg, N=227 | 43.6
  8 weeks: <120 mm Hg, N=227 | 18.1
  12 weeks: <140 mm Hg, N=227 | 80.6
  12 weeks: <135 mm Hg, N=227 | 70.0
  12 weeks: <130 mm Hg, N=227 | 56.8
  12 weeks: <120 mm Hg, N=227 | 28.6
  16 weeks: <140 mm Hg, N=227 | 87.7
  16 weeks: <135 mm Hg, N=227 | 79.7
  16 weeks: <130 mm Hg, N=227 | 70.9
  16 weeks: <120 mm Hg, N=227 | 43.6
  20 weeks: <140 mm Hg, N=227 | 91.6
  20 weeks: <135 mm Hg, N=227 | 85.9
  20 weeks: <130 mm Hg, N=227 | 78.9
  20 weeks: <120 mm Hg, N=227 | 50.7

33. Secondary Outcome: Percentage of Elderly Patients Achieving Seated Diastolic Blood Pressure Goal From Baseline to 4, 8, 12, 16, 20 Weeks
Time Frame: Baseline to 4, 8, 12, 16, 20 weeks
Population: The analysis population consists of those elderly participants who have a baseline and at least 1 post-baseline measurement and who received at least one dose of study medication. However, the number of participants included will vary because of missing data and the number of dropouts. Elderly is defined as greater than or = to 65 years of age.
Measure: Number; unit: Percentage of Participants
Arm/Group | Olmesartan Medoxomil/Amlodipine Tablets + Hydrochlorothiazide
Number analyzed (Participants) | 227
Percentage of Participants
  4 weeks: <90 mm Hg, N=227 | 88.1
  4 weeks: <85 mm Hg, N=227 | 76.7
  4 weeks: <80 mm Hg, N=227 | 58.2
  8 weeks: <90 mm Hg, N=227 | 92.1
  8 weeks: <85 mm Hg, N=227 | 83.7
  8 weeks: <80 mm Hg, N=227 | 71.8
  12 weeks: <90 mm Hg, N=227 | 97.4
  12 weeks: <85 mm Hg, N=227 | 92.1
  12 weeks: <80 mm Hg, N=227 | 80.2
  16 weeks: <90 mm Hg, N=227 | 98.7
  16 weeks: <85 mm Hg, N=227 | 94.3
  16 weeks: <80 mm Hg, N=227 | 88.6
  20 weeks: <90 mm Hg, N=227 | 98.7
  20 weeks: <85 mm Hg, N=227 | 95.2
  20 weeks: <80 mm Hg, N=227 | 90.3

34. Secondary Outcome: Percentage of Elderly Patients Achieving Seated Systolic Blood Pressure Reduction Ranges From Baseline to 4, 8, 12, 16, 20 Weeks
Time Frame: Baseline to 4, 8, 12, 16, 20 weeks
Population: as for outcome 33
Measure: Number; unit: Percentage of Participants
Arm/Group | Olmesartan Medoxomil/Amlodipine Tablets + Hydrochlorothiazide
Number analyzed (Participants) | 224
Percentage of Participants
  4 weeks: ≤ 15 mm Hg, N=224 | 47.3
  4 weeks: >15 and ≤ 30 mm Hg, N=224 | 40.2
  4 weeks: >30 and ≤ 45 mm Hg, N=224 | 11.2
  4 weeks: >45 mm Hg, N=224 | 1.3
  8 weeks: ≤ 15 mm Hg, N=217 | 42.9
  8 weeks: >15 and ≤ 30 mm Hg, N=217 | 37.8
  8 weeks: >30 and ≤ 45 mm Hg, N=217 | 16.6
  8 weeks: >45 mm Hg, N=217 | 2.8
  12 weeks: ≤ 15 mm Hg, N=199 | 26.6
  12 weeks: >15 and ≤ 30 mm Hg, N=199 | 46.7
  12 weeks: >30 and ≤ 45 mm Hg, N=199 | 24.6
  12 weeks: >45 mm Hg, N=199 | 2.0
  16 weeks: ≤ 15 mm Hg, N=179 | 17.9
  16 weeks: >15 and ≤ 30 mm Hg, N=179 | 32.4
  16 weeks: >30 and ≤ 45 mm Hg, N=179 | 39.7
  16 weeks: >45 mm Hg, N=179 | 10.1
  20 weeks: ≤ 15 mm Hg, N=166 | 14.5
  20 weeks: >15 and ≤ 30 mm Hg, N=166 | 37.4
  20 weeks: >30 and ≤ 45 mm Hg, N=166 | 38.0
  20 weeks: >45 mm Hg, N=166 | 10.2

35. Secondary Outcome: Percentage of Elderly Patients Achieving Seated Diastolic Blood Pressure Reduction Ranges From Baseline to 4, 8, 12, 16, 20 Weeks
Time Frame: Baseline to 4, 8, 12, 16, 20 weeks
Population: as for outcome 33
Measure: Number; unit: Percentage of Participants
Arm/Group | Olmesartan Medoxomil/Amlodipine Tablets + Hydrochlorothiazide
Number analyzed (Participants) | 224
Percentage of Participants
  4 weeks: ≤ 10 mm Hg, N=224 | 63.8
  4 weeks: >10 and ≤ 15 mm Hg, N=224 | 20.5
  4 weeks: >15 and ≤ 20 mm Hg, N=224 | 9.4
  4 weeks: >20 mm Hg, N=224 | 6.3
  8 weeks: ≤ 10 mm Hg, N=217 | 57.1
  8 weeks: >10 and ≤ 15 mm Hg, N=217 | 19.8
  8 weeks: >15 and ≤ 20 mm Hg, N=217 | 14.3
  8 weeks: >20 mm Hg, N=217 | 8.8
  12 weeks: ≤ 10 mm Hg, N=199 | 45.2
  12 weeks: >10 and ≤15 mm Hg, N=199 | 25.1
  12 weeks: >15 and ≤ 20 mm Hg, N=199 | 15.6
  12 weeks: >20 mm Hg, N=199 | 14.1
  16 weeks: ≤ 10 mm Hg, N=179 | 27.4
  16 weeks: >10 and ≤ 15 mm Hg, N=179 | 25.1
  16 weeks: >15 and ≤ 20 mm Hg, N=179 | 22.9
  16 weeks: >20 mm Hg, N=179 | 24.6
  20 weeks: ≤ 10 mm Hg, N=166 | 34.9
  20 weeks: >10 and ≤ 15 mm Hg, N=166 | 20.5
  20 weeks: >15 and ≤ 20 mm Hg, N=166 | 24.1
  20 weeks: >20 mm Hg, N=166 | 20.5

36. Secondary Outcome: Percentage of Type 2 Diabetic Patients Achieving Seated Systolic Blood Pressure Goal From Baseline to 4, 8, 12, 16, 20 Weeks
Time Frame: Baseline to 4, 8, 12, 16, 20 weeks
Population: The analysis population consists of those type 2 diabetic participants who have a baseline and at least 1 post-baseline measurement and who received at least one dose of study medication. However, the number of participants included may vary because of missing data and the number of dropouts.
Measure: Number; unit: Percentage of Participants
Arm/Group | Olmesartan Medoxomil/Amlodipine Tablets + Hydrochlorothiazide
Number analyzed (Participants) | 190
Percentage of Participants
  4 weeks: <140 mm Hg, N=190 | 54.7
  4 weeks: <135 mm Hg, N=190 | 41.1
  4 weeks: <130 mm Hg, N=190 | 26.3
  4 weeks: <120 mm Hg, N=190 | 10.0
  8 weeks: <140 mm Hg, N=190 | 69.0
  8 weeks: <135 mm Hg, N=190 | 56.3
  8 weeks: <130 mm Hg, N=190 | 42.6
  8 weeks: <120 mm Hg, N=190 | 15.8
  12 weeks: <140 mm Hg, N=190 | 81.6
  12 weeks: <135 mm Hg, N=190 | 69.5
  12 weeks: <130 mm Hg, N=190 | 57.9
  12 weeks: <120 mm Hg, N=190 | 30.0
  16 weeks: <140 mm Hg, N=190 | 87.9
  16 weeks: <135 mm Hg, N=190 | 79.0
  16 weeks: <130 mm Hg, N=190 | 69.0
  16 weeks: <120 mm Hg, N=190 | 39.5
  20 weeks: <140 mm Hg, N=190 | 91.1
  20 weeks: <135 mm Hg, N=190 | 84.2
  20 weeks: <130 mm Hg, N=190 | 75.3
  20 weeks: <120 mm Hg, N=190 | 48.4

37. Secondary Outcome: Percentage of Type 2 Diabetic Patients Achieving Seated Diastolic Blood Pressure Goal From Baseline to 4, 8, 12, 16, 20 Weeks
Time Frame: Baseline to 4, 8, 12, 16, 20 weeks
Population: as for outcome 36
Measure: Number; unit: Percentage of Participants
Arm/Group | Olmesartan Medoxomil/Amlodipine Tablets + Hydrochlorothiazide
Number analyzed (Participants) | 190
Percentage of Participants
  4 weeks: <90 mm Hg, N=190 | 75.8
  4 weeks: <85 mm Hg, N=190 | 64.2
  4 weeks: <80 mm Hg, N=190 | 39.0
  8 weeks: <90 mm Hg, N=190 | 85.8
  8 weeks: <85 mm Hg, N=190 | 72.6
  8 weeks: <80 mm Hg, N=190 | 51.1
  12 weeks: <90 mm Hg, N=190 | 94.2
  12 weeks: <85 mm Hg, N=190 | 83.2
  12 weeks: <80 mm Hg, N=190 | 63.7
  16 weeks: <90 mm Hg, N=190 | 97.9
  16 weeks: <85 mm Hg, N=190 | 89.0
  16 weeks: <80 mm Hg, N=190 | 70.5
  20 weeks: <90 mm Hg, N=190 | 99.0
  20 weeks: <85 mm Hg, N=190 | 90.5
  20 weeks: <80 mm Hg, N=190 | 76.8

38. Secondary Outcome: Percentage of Type 2 Diabetic Patients Achieving Seated Systolic Blood Pressure Reduction Ranges From Baseline to 4, 8, 12, 16, 20 Weeks
Time Frame: Baseline to 4, 8, 12, 16, 20 weeks
Population: as for outcome 36
Measure: Number; unit: Percentage of Participants
Arm/Group | Olmesartan Medoxomil/Amlodipine Tablets + Hydrochlorothiazide
Number analyzed (Participants) | 189
Percentage of Participants
  4 weeks: ≤ 15 mm Hg, N=189 | 56.1
  4 weeks: >15 and ≤ 30 mm Hg, N=189 | 36.0
  4 weeks: >30 and ≤ 45 mm Hg, N=189 | 7.9
  4 weeks: >45 mm Hg, N=189 | 0.0
  8 weeks: ≤ 15 mm Hg, N=181 | 54.1
  8 weeks: >15 and ≤ 30 mm Hg, N=181 | 34.3
  8 weeks: >30 and ≤ 45 mm Hg, N=181 | 11.6
  8 weeks: >45 mm Hg, N=181 | 0.0
  12 weeks: ≤ 15 mm Hg, N=170 | 35.3
  12 weeks: >15 and ≤ 30 mm Hg, N=170 | 38.2
  12 weeks: >30 and ≤ 45 mm Hg, N=170 | 22.9
  12 weeks: >45 mm Hg, N=170 | 3.5
  16 weeks: ≤ 15 mm Hg, N=156 | 28.2
  16 weeks: >15 and ≤ 30 mm Hg, N=156 | 40.4
  16 weeks: >30 and ≤ 45 mm Hg, N=156 | 26.3
  16 weeks: >45 mm Hg, N=156 | 5.1
  20 weeks: ≤ 15 mm Hg, N=150 | 26.0
  20 weeks: >15 and ≤ 30 mm Hg, N=150 | 40.0
  20 weeks: >30 and ≤ 45 mm Hg, N=150 | 26.7
  20 weeks: >45 mm Hg, N=150 | 7.3

39. Secondary Outcome: Percentage of Type 2 Diabetic Patients Achieving Seated Diastolic Blood Pressure Reduction Ranges From Baseline to 4, 8, 12, 16, 20 Weeks
Time Frame: Baseline to 4, 8, 12, 16, 20 weeks
Population: The analysis population consists of those type 2 diabetic participants who have a baseline and at least 1 post-baseline measurement and who received at least one dose of study medication. However, the number of participants included will vary because of missing data and the number of dropouts.
Measure: Number; unit: Percentage of Participants
Arm/Group | Olmesartan Medoxomil/Amlodipine Tablets + Hydrochlorothiazide
Number analyzed (Participants) | 189
Percentage of Participants
  4 weeks: ≤ 10 mm Hg, N=189 | 67.7
  4 weeks: >10 and ≤ 15 mm Hg, N=189 | 16.9
  4 weeks: >15 and ≤ 20 mm Hg, N=189 | 11.6
  4 weeks: >20 mm Hg, N=189 | 3.7
  8 weeks: ≤ 10 mm Hg, N=181 | 60.8
  8 weeks: >10 and ≤ 15 mm Hg, N=181 | 20.4
  8 weeks: >15 and ≤ 20 mm Hg, N=181 | 14.9
  8 weeks: >20 mm Hg, N=181 | 3.9
  12 weeks: ≤ 10 mm Hg, N=170 | 41.2
  12 weeks: >10 and ≤15 mm Hg, N=170 | 32.4
  12 weeks: >15 and ≤ 20 mm Hg, N=170 | 12.9
  12 weeks: >20 mm Hg, N=170 | 13.5
  16 weeks: ≤ 10 mm Hg, N=156 | 32.7
  16 weeks: >10 and ≤ 15 mm Hg, N=156 | 26.9
  16 weeks: >15 and ≤ 20 mm Hg, N=156 | 21.8
  16 weeks: >20 mm Hg, N=156 | 18.6
  20 weeks: ≤ 10 mm Hg, N=150 | 37.3
  20 weeks: >10 and ≤ 15 mm Hg, N=150 | 18.0
  20 weeks: >15 and ≤ 20 mm Hg, N=150 | 26.0
  20 weeks: >20 mm Hg, N=150 | 18.7

40. Secondary Outcome: Percentage of Obese Patients Achieving Seated Systolic Blood Pressure Goal From Baseline to 4, 8, 12, 16, 20 Weeks
Time Frame: Baseline to 4, 8, 12, 16, 20 weeks
Population: The analysis population consists of those obese participants who have a baseline and at least 1 post-baseline measurement and who received at least one dose of study medication. However, the number of participants included may vary because of missing data and the number of dropouts. Obesity is defined as Body Mass Index ≥30 kg/m2
Measure: Number; unit: Percentage of Participants
Arm/Group | Olmesartan Medoxomil/Amlodipine Tablets + Hydrochlorothiazide
Number analyzed (Participants) | 497
Percentage of Participants
  4 weeks: <140 mm Hg, N=497 | 51.3
  4 weeks: <135 mm Hg, N=497 | 37.2
  4 weeks: <130 mm Hg, N=497 | 23.3
  4 weeks: <120 mm Hg, N=497 | 7.9
  8 weeks: <140 mm Hg, N=500 | 63.2
  8 weeks: <135 mm Hg, N=500 | 49.2
  8 weeks: <130 mm Hg, N=500 | 37.0
  8 weeks: <120 mm Hg, N=500 | 13.8
  12 weeks: <140 mm Hg, N=500 | 76.6
  12 weeks: <135 mm Hg, N=500 | 61.6
  12 weeks: <130 mm Hg, N=500 | 49.2
  12 weeks: <120 mm Hg, N=500 | 23.2
  16 weeks: <140 mm Hg, N=500 | 85.8
  16 weeks: <135 mm Hg, N=500 | 75.6
  16 weeks: <130 mm Hg, N=500 | 63.6
  16 weeks: <120 mm Hg, N=500 | 34.6
  20 weeks: <140 mm Hg, N=500 | 90.2
  20 weeks: <135 mm Hg, N=500 | 82.6
  20 weeks: <130 mm Hg, N=500 | 72.2
  20 weeks: <120 mm Hg, N=500 | 43.0

41. Secondary Outcome: Percentage of Obese Patients Achieving Seated Diastolic Blood Pressure Goal From Baseline to 4, 8, 12, 16, 20 Weeks
Time Frame: Baseline to 4, 8, 12, 16, 20 weeks
Population: as for outcome 40
Measure: Number; unit: Percentage of Participants
Arm/Group | Olmesartan Medoxomil/Amlodipine Tablets + Hydrochlorothiazide
Number analyzed (Participants) | 497
Percentage of Participants
  4 weeks: <90 mm Hg, N=497 | 63.2
  4 weeks: <85 mm Hg, N=497 | 46.3
  4 weeks: <80 mm Hg, N=497 | 26.0
  8 weeks: <90 mm Hg, N=497 | 77.2
  8 weeks: <85 mm Hg, N=500 | 59.4
  8 weeks: <80 mm Hg, N=500 | 38.8
  12 weeks: <90 mm Hg, N=500 | 86.6
  12 weeks: <85 mm Hg, N=500 | 69.8
  12 weeks: <80 mm Hg, N=500 | 48.4
  16 weeks: <90 mm Hg, N=500 | 93.2
  16 weeks: <85 mm Hg, N=500 | 80.4
  16 weeks: <80 mm Hg, N=500 | 60.4
  20 weeks: <90 mm Hg, N=500 | 94.6
  20 weeks: <85 mm Hg, N=500 | 83.8
  20 weeks: <80 mm Hg, N=500 | 67.6

42. Secondary Outcome: Percentage of Obese Patients Achieving Seated Systolic Blood Pressure Reduction Ranges From Baseline to 4, 8, 12, 16, 20 Weeks
Time Frame: Baseline to 4, 8, 12, 16, 20 weeks
Population: as for outcome 40
Measure: Number; unit: Percentage of Participants
Arm/Group | Olmesartan Medoxomil/Amlodipine Tablets + Hydrochlorothiazide
Number analyzed (Participants) | 495
Percentage of Participants
  4 weeks: ≤ 15 mm Hg, N=495 | 56.0
  4 weeks: >15 and ≤ 30 mm Hg, N=495 | 35.2
  4 weeks: >30 and ≤ 45 mm Hg, N=495 | 8.5
  4 weeks: >45 mm Hg, N=495 | 0.4
  8 weeks: ≤ 15 mm Hg, N=468 | 52.4
  8 weeks: >15 and ≤ 30 mm Hg, N=468 | 35.9
  8 weeks: >30 and ≤ 45 mm Hg, N=468 | 10.3
  8 weeks: >45 mm Hg, N=468 | 1.5
  12 weeks: ≤ 15 mm Hg, N=436 | 37.8
  12 weeks: >15 and ≤ 30 mm Hg, N=436 | 42.4
  12 weeks: >30 and ≤ 45 mm Hg, N=436 | 17.4
  12 weeks: >45 mm Hg, N=436 | 2.5
  16 weeks: ≤ 15 mm Hg, N=400 | 27.8
  16 weeks: >15 and ≤ 30 mm Hg, N=400 | 36.0
  16 weeks: >30 and ≤ 45 mm Hg, N=400 | 27.5
  16 weeks: >45 mm Hg, N=400 | 8.8
  20 weeks: ≤ 15 mm Hg, N=379 | 20.6
  20 weeks: >15 and ≤ 30 mm Hg, N=379 | 37.5
  20 weeks: >30 and ≤ 45 mm Hg, N=379 | 33.3
  20 weeks: >45 mm Hg, N=379 | 8.7

43. Secondary Outcome: Percentage of Obese Patients Achieving Seated Diastolic Blood Pressure Reduction Ranges From Baseline to 4, 8, 12, 16, 20 Weeks
Time Frame: Baseline to 4, 8, 12, 16, 20 weeks
Population: The analysis population consists of those obese participants who have a baseline and at least 1 post-baseline measurement and who received at least one dose of study medication. However, the number of participants included will vary because of missing data and the number of dropouts. Obesity is defined as Body Mass Index ≥30 kg/m2
Measure: Number; unit: Percentage of Participants
Arm/Group | Olmesartan Medoxomil/Amlodipine Tablets + Hydrochlorothiazide
Number analyzed (Participants) | 495
Percentage of Participants
  4 weeks: ≤ 10 mm Hg, N=495 | 67.5
  4 weeks: >10 and ≤ 15 mm Hg, N=495 | 17.8
  4 weeks: >15 and ≤ 20 mm Hg, N=495 | 8.5
  4 weeks: >20 mm Hg, N=495 | 6.3
  8 weeks: ≤ 10 mm Hg, N=468 | 59.4
  8 weeks: >10 and ≤ 15 mm Hg, N=468 | 19.9
  8 weeks: >15 and ≤ 20 mm Hg, N=468 | 13.0
  8 weeks: >20 mm Hg, N=468 | 7.7
  12 weeks: ≤ 10 mm Hg, N=436 | 48.9
  12 weeks: >10 and ≤15 mm Hg, N=436 | 22.5
  12 weeks: >15 and ≤ 20 mm Hg, N=436 | 16.1
  12 weeks: >20 mm Hg, N=436 | 12.6
  16 weeks: ≤ 10 mm Hg, N=400 | 33.3
  16 weeks: >10 and ≤ 15 mm Hg, N=400 | 23.0
  16 weeks: >15 and ≤ 20 mm Hg, N=400 | 19.0
  16 weeks: >20 mm Hg, N=400 | 24.8
  20 weeks: ≤ 10 mm Hg, N=379 | 31.9
  20 weeks: >10 and ≤ 15 mm Hg, N=379 | 18.7
  20 weeks: >15 and ≤ 20 mm Hg, N=379 | 22.4
  20 weeks: >20 mm Hg, N=379 | 26.9

44. Secondary Outcome: Percentage of Patients With Metabolic Syndrome Achieving Seated Systolic Blood Pressure Goal From Baseline to 4, 8, 12, 16, 20 Weeks
Time Frame: Baseline to 4, 8, 12, 16, 20 weeks
Population: Subjects with metabolic syndrome (MS) who have a baseline and at least 1 post-baseline measurement and who received at least one dose of study medication. The number may vary due to missing data and the number of dropouts. MS is defined using waist size,and triglyceride, cholesterol, blood pressure, and body mass index values.
Measure: Number; unit: Percentage of Participants
Arm/Group | Olmesartan Medoxomil/Amlodipine Tablets + Hydrochlorothiazide
Number analyzed (Participants) | 454
Percentage of Participants
  4 weeks: <140 mm Hg, N=454 | 56.4
  4 weeks: <135 mm Hg, N=454 | 41.4
  4 weeks: <130 mm Hg, N=454 | 27.1
  4 weeks: <120 mm Hg, N=454 | 7.9
  8 weeks: <140 mm Hg, N=457 | 67.6
  8 weeks: <135 mm Hg, N=457 | 54.3
  8 weeks: <130 mm Hg, N=457 | 40.9
  8 weeks: <120 mm Hg, N=457 | 16.2
  12 weeks: <140 mm Hg, N=457 | 81.4
  12 weeks: <135 mm Hg, N=457 | 67.2
  12 weeks: <130 mm Hg, N=457 | 54.1
  12 weeks: <120 mm Hg, N=457 | 27.6
  16 weeks: <140 mm Hg, N=457 | 88.8
  16 weeks: <135 mm Hg, N=457 | 80.3
  16 weeks: <130 mm Hg, N=457 | 67.0
  16 weeks: <120 mm Hg, N=457 | 39.0
  20 weeks: <140 mm Hg, N=457 | 91.5
  20 weeks: <135 mm Hg, N=457 | 85.6
  20 weeks: <130 mm Hg, N=457 | 74.8
  20 weeks: <120 mm Hg, N=457 | 47.1

45. Secondary Outcome: Percentage of Patients With Metabolic Syndrome Achieving Seated Diastolic Blood Pressure Goal From Baseline to 4, 8, 12, 16, 20 Weeks
Time Frame: Baseline to 4, 8, 12, 16, 20 weeks
Population: as for outcome 44
Measure: Number; unit: Percentage of Participants
Arm/Group | Olmesartan Medoxomil/Amlodipine Tablets + Hydrochlorothiazide
Number analyzed (Participants) | 454
Percentage of Participants
  4 weeks: <90 mm Hg, N=454 | 69.6
  4 weeks: <85 mm Hg, N=454 | 53.5
  4 weeks: <80 mm Hg, N=454 | 31.9
  8 weeks: <90 mm Hg, N=457 | 82.1
  8 weeks: <85 mm Hg, N=457 | 66.1
  8 weeks: <80 mm Hg, N=457 | 43.5
  12 weeks: <90 mm Hg, N=457 | 90.4
  12 weeks: <85 mm Hg, N=457 | 76.6
  12 weeks: <80 mm Hg, N=457 | 56.5
  16 weeks: <90 mm Hg, N=457 | 94.8
  16 weeks: <85 mm Hg, N=457 | 83.2
  16 weeks: <80 mm Hg, N=457 | 65.9
  20 weeks: <90 mm Hg, N=457 | 95.4
  20 weeks: <85 mm Hg, N=457 | 86.2
  20 weeks: <80 mm Hg, N=457 | 72.0

46. Secondary Outcome: Percentage of Patients With Metabolic Syndrome Achieving Seated Systolic Blood Pressure Reduction Ranges From Baseline to 4, 8, 12, 16, 20 Weeks
Time Frame: Baseline to 4, 8, 12, 16, 20 weeks
Population: as for outcome 44
Measure: Number; unit: Percentage of Participants
Arm/Group | Olmesartan Medoxomil/Amlodipine Tablets + Hydrochlorothiazide
Number analyzed (Participants) | 453
Percentage of Participants
  4 weeks: ≤ 15 mm Hg, N=453 | 49.5
  4 weeks: >15 and ≤ 30 mm Hg, N=453 | 38.4
  4 weeks: >30 and ≤ 45 mm Hg, N=453 | 11.5
  4 weeks: >45 mm Hg, N=453 | 0.7
  8 weeks: ≤ 15 mm Hg, N=431 | 48.0
  8 weeks: >15 and ≤ 30 mm Hg, N=431 | 35.5
  8 weeks: >30 and ≤ 45 mm Hg, N=431 | 14.4
  8 weeks: >45 mm Hg, N=431 | 2.1
  12 weeks: ≤ 15 mm Hg, N=402 | 30.4
  12 weeks: >15 and ≤ 30 mm Hg, N=402 | 43.8
  12 weeks: >30 and ≤ 45 mm Hg, N=402 | 22.6
  12 weeks: >45 mm Hg, N=402 | 3.2
  16 weeks: ≤ 15 mm Hg, N=371 | 24.0
  16 weeks: >15 and ≤ 30 mm Hg, N=371 | 37.7
  16 weeks: >30 and ≤ 45 mm Hg, N=371 | 29.1
  16 weeks: >45 mm Hg, N=371 | 9.2
  20 weeks: ≤ 15 mm Hg, N=356 | 19.7
  20 weeks: >15 and ≤ 30 mm Hg, N=356 | 36.5
  20 weeks: >30 and ≤ 45 mm Hg, N=356 | 36.0
  20 weeks: >45 mm Hg, N=356 | 7.9

47. Secondary Outcome: Percentage of Patients With Metabolic Syndrome Achieving Seated Diastolic Blood Pressure Reduction Ranges From Baseline to 4, 8, 12, 16, 20 Weeks
Time Frame: Baseline to 4, 8, 12, 16, 20 weeks
Population: as for outcome 44
Measure: Number; unit: Percentage of Participants
Arm/Group | Olmesartan Medoxomil/Amlodipine Tablets + Hydrochlorothiazide
Number analyzed (Participants) | 453
Percentage of Participants
  4 weeks: ≤ 10 mm Hg, N=453 | 62.7
  4 weeks: >10 and ≤ 15 mm Hg, N=453 | 22.3
  4 weeks: >15 and ≤ 20 mm Hg, N=453 | 8.6
  4 weeks: >20 mm Hg, N=453 | 6.4
  8 weeks: ≤ 10 mm Hg, N=431 | 56.6
  8 weeks: >10 and ≤ 15 mm Hg, N=431 | 19.7
  8 weeks: >15 and ≤ 20 mm Hg, N=431 | 15.3
  8 weeks: >20 mm Hg, N=431 | 8.4
  12 weeks: ≤ 10 mm Hg, N=402 | 44.3
  12 weeks: >10 and ≤15 mm Hg, N=402 | 22.1
  12 weeks: >15 and ≤ 20 mm Hg, N=402 | 17.4
  12 weeks: >20 mm Hg, N=402 | 16.2
  16 weeks: ≤ 10 mm Hg, N=371 | 32.4
  16 weeks: >10 and ≤ 15 mm Hg, N=371 | 24.0
  16 weeks: >15 and ≤ 20 mm Hg, N=371 | 21.0
  16 weeks: >20 mm Hg, N=371 | 22.6
  20 weeks: ≤ 10 mm Hg, N=356 | 33.2
  20 weeks: >10 and ≤ 15 mm Hg, N=356 | 19.4
  20 weeks: >15 and ≤ 20 mm Hg, N=356 | 22.5
  20 weeks: >20 mm Hg, N=356 | 25.0

48. Secondary Outcome: Percentage of Participants Previously on a Dihydropyridine Calcium Channel Blocker Achieving the Blood Pressure Goals From Baseline to 12 Weeks
Time Frame: Baseline to 12 weeks
Population: Participants previously on a Dihydropyridine Calcium Channel Blocker who have received at least one dose of study medication and who have a baseline value.
Measure: Number; unit: Percentage of participants
Arm/Group | Olmesartan Medoxomil/Amlodipine Tablets + Hydrochlorothiazide
Number analyzed (Participants) | 117
Percentage of participants
  Systolic blood pressure <140 mmHg | 73.5
  Systolic blood pressure <135 mmHg | 59.0
  Systolic blood pressure <130 mmHg | 47.9
  Systolic blood pressure <120 mmHg | 18.8
  Diastolic blood pressure <90 mmHg | 86.3
  Diastolic blood pressure <85 mmHg | 72.7
  Diastolic blood pressure <80 mmHg | 48.7
  Blood pressure <140/90 mmHg | 68.4
  Blood pressure <135/80 mmHg | 40.2
  Blood pressure <130/80 mmHg | 34.2
  Blood pressure <120/80 mmHg | 16.2

49. Secondary Outcome: Percentage of Participants Previously on a Dihydropyridine Calcium Channel Blocker Achieving the Blood Pressure Goals From Baseline to 20 Weeks
Time Frame: Baseline to 20 weeks
Population: as for outcome 48
Measure: Number; unit: Percentage of participants
Arm/Group | Olmesartan Medoxomil/Amlodipine Tablets + Hydrochlorothiazide
Number analyzed (Participants) | 117
Percentage of participants
  Systolic blood pressure <140 mmHg | 89.7
  Systolic blood pressure <135 mmHg | 83.8
  Systolic blood pressure <130 mmHg | 69.2
  Systolic blood pressure <120 mmHg | 41.0
  Diastolic blood pressure <90 mmHg | 91.5
  Diastolic blood pressure <85 mmHg | 85.5
  Diastolic blood pressure <80 mmHg | 69.2
  Blood pressure <140/90 mmHg | 85.5
  Blood pressure <135/80 mmHg | 64.1
  Blood pressure <130/80 mmHg | 59.8
  Blood pressure <120/80 mmHg | 36.8

50. Secondary Outcome: Percentage of Participants Previously on a Diuretic Achieving the Blood Pressure Goals From Baseline to 12 Weeks
Time Frame: Baseline to 12 weeks
Population: Participants previously on a diuretic who have received at least one dose of study medication and who have a baseline value.
Measure: Number; unit: Percentage of participants
Arm/Group | Olmesartan Medoxomil/Amlodipine Tablets + Hydrochlorothiazide
Number analyzed (Participants) | 166
Percentage of participants
  Systolic blood pressure <140 mmHg | 92.8
  Systolic blood pressure <135 mmHg | 82.5
  Systolic blood pressure <130 mmHg | 78.3
  Systolic blood pressure <120 mmHg | 51.2
  Diastolic blood pressure <90 mmHg | 94.6
  Diastolic blood pressure <85 mmHg | 86.8
  Diastolic blood pressure <80 mmHg | 71.7
  Blood pressure <140/90 mmHg | 88.6
  Blood pressure <135/80 mmHg | 67.5
  Blood pressure <130/80 mmHg | 65.1
  Blood pressure <120/80 mmHg | 48.2

51. Secondary Outcome: Percentage of Participants Previously on a Diuretic Achieving the Blood Pressure Goals From Baseline to 20 Weeks
Time Frame: Baseline to 20 weeks
Population: as for outcome 50
Measure: Number; unit: Percentage of participants
Arm/Group | Olmesartan Medoxomil/Amlodipine Tablets + Hydrochlorothiazide
Number analyzed (Participants) | 166
Percentage of participants
  Systolic blood pressure <140 mmHg | 92.8
  Systolic blood pressure <135 mmHg | 82.5
  Systolic blood pressure <130 mmHg | 78.3
  Systolic blood pressure <120 mmHg | 51.2
  Diastolic blood pressure <90 mmHg | 94.6
  Diastolic blood pressure <85 mmHg | 86.8
  Diastolic blood pressure <80 mmHg | 71.7
  Blood pressure <140/90 mmHg | 88.6
  Blood pressure <135/80 mmHg | 67.5
  Blood pressure <130/80 mmHg | 65.1
  Blood pressure <120/80 mmHg | 48.2

52. Secondary Outcome: Percentage of Participants Previously on an Angiotensin Converting Enzyme Inhibitor Achieving the Blood Pressure Goals From Baseline to 12 Weeks
Time Frame: Baseline to 12 weeks
Population: Participants previously on an angiotensin converting enzyme inhibitor who have received at least one dose of study medication and who have a baseline value.
Measure: Number; unit: Percentage of participants
Arm/Group | Olmesartan Medoxomil/Amlodipine Tablets + Hydrochlorothiazide
Number analyzed (Participants) | 283
Percentage of participants
  Systolic blood pressure <140 mmHg | 81.3
  Systolic blood pressure <135 mmHg | 69.3
  Systolic blood pressure <130 mmHg | 53.0
  Systolic blood pressure <120 mmHg | 31.5
  Diastolic blood pressure <90 mmHg | 94.4
  Diastolic blood pressure <85 mmHg | 80.6
  Diastolic blood pressure <80 mmHg | 64.3
  Blood pressure <140/90 mmHg | 78.5
  Blood pressure <135/80 mmHg | 52.7
  Blood pressure <130/80 mmHg | 43.5
  Blood pressure <120/80 mmHg | 27.9

53. Secondary Outcome: Percentage of Participants Previously on an Angiotensin Converting Enzyme Inhibitor Achieving the Blood Pressure Goals From Baseline to 20 Weeks
Time Frame: Baseline to 20 weeks
Population: as for outcome 52
Measure: Number; unit: Percentage of participants
Arm/Group | Olmesartan Medoxomil/Amlodipine Tablets + Hydrochlorothiazide
Number analyzed (Participants) | 283
Percentage of participants
  Systolic blood pressure <140 mmHg | 91.5
  Systolic blood pressure <135 mmHg | 84.5
  Systolic blood pressure <130 mmHg | 71.4
  Systolic blood pressure <120 mmHg | 47.4
  Diastolic blood pressure <90 mmHg | 98.2
  Diastolic blood pressure <85 mmHg | 89.8
  Diastolic blood pressure <80 mmHg | 78.5
  Blood pressure <140/90 mmHg | 90.5
  Blood pressure <135/80 mmHg | 71.0
  Blood pressure <130/80 mmHg | 61.5
  Blood pressure <120/80 mmHg | 44.5

54. Secondary Outcome: Percentage of Participants Previously on an Angiotensin II Receptor Blocker Achieving the Blood Pressure Goals From Baseline to 12 Weeks
Time Frame: Baseline to 12 weeks
Population: Participants previously on an angiotensin II receptor blocker who have received at least one dose of study medication and who have a baseline value.
Measure: Number; unit: Percentage of participants
Arm/Group | Olmesartan Medoxomil/Amlodipine Tablets + Hydrochlorothiazide
Number analyzed (Participants) | 234
Percentage of participants
  Systolic blood pressure <140 mmHg | 80.8
  Systolic blood pressure <135 mmHg | 69.2
  Systolic blood pressure <130 mmHg | 56.0
  Systolic blood pressure <120 mmHg | 26.1
  Diastolic blood pressure <90 mmHg | 89.7
  Diastolic blood pressure <85 mmHg | 76.9
  Diastolic blood pressure <80 mmHg | 59.0
  Blood pressure <140/90 mmHg | 76.1
  Blood pressure <135/80 mmHg | 52.6
  Blood pressure <130/80 mmHg | 46.2
  Blood pressure <120/80 mmHg | 23.1

55. Secondary Outcome: Percentage of Participants Previously on an Angiotensin II Receptor Blocker Achieving the Blood Pressure Goals From Baseline to 20 Weeks
Time Frame: Baseline to 20 weeks
Population: as for outcome 54
Measure: Number; unit: Percentage of participants
Arm/Group | Olmesartan Medoxomil/Amlodipine Tablets + Hydrochlorothiazide
Number analyzed (Participants) | 234
Percentage of participants
  Systolic blood pressure <140 mmHg | 92.3
  Systolic blood pressure <135 mmHg | 87.2
  Systolic blood pressure <130 mmHg | 79.5
  Systolic blood pressure <120 mmHg | 47.4
  Diastolic blood pressure <90 mmHg | 96.6
  Diastolic blood pressure <85 mmHg | 89.3
  Diastolic blood pressure <80 mmHg | 74.8
  Blood pressure <140/90 mmHg | 90.6
  Blood pressure <135/80 mmHg | 70.1
  Blood pressure <130/80 mmHg | 65.0
  Blood pressure <120/80 mmHg | 44.0

56. Secondary Outcome: Percentage of Participants Previously on a Beta Blocker Achieving the Blood Pressure Goals From Baseline to 12 Weeks
Time Frame: Baseline to 12 weeks
Population: Participants previously on an beta blocker who have received at least one dose of study medication and who have a baseline value.
Measure: Number; unit: Percentage of participants
Arm/Group | Olmesartan Medoxomil/Amlodipine Tablets + Hydrochlorothiazide
Number analyzed (Participants) | 113
Percentage of participants
  Systolic blood pressure <140 mmHg | 88.5
  Systolic blood pressure <135 mmHg | 75.2
  Systolic blood pressure <130 mmHg | 62.0
  Systolic blood pressure <120 mmHg | 33.6
  Diastolic blood pressure <90 mmHg | 94.7
  Diastolic blood pressure <85 mmHg | 83.2
  Diastolic blood pressure <80 mmHg | 61.1
  Blood pressure <140/90 mmHg | 86.7
  Blood pressure <135/80 mmHg | 55.8
  Blood pressure <130/80 mmHg | 49.6
  Blood pressure <120/80 mmHg | 29.2

57. Secondary Outcome: Percentage of Participants Previously on a Beta Blocker Achieving the Blood Pressure Goals From Baseline to 20 Weeks
Time Frame: Baseline to 20 weeks
Population: as for outcome 56
Measure: Number; unit: Percentage of participants
Arm/Group | Olmesartan Medoxomil/Amlodipine Tablets + Hydrochlorothiazide
Number analyzed (Participants) | 113
Percentage of participants
  Systolic blood pressure <140 mmHg | 93.8
  Systolic blood pressure <135 mmHg | 87.6
  Systolic blood pressure <130 mmHg | 79.7
  Systolic blood pressure <120 mmHg | 47.8
  Diastolic blood pressure <90 mmHg | 98.2
  Diastolic blood pressure <85 mmHg | 89.4
  Diastolic blood pressure <80 mmHg | 77.0
  Blood pressure <140/90 mmHg | 92.9
  Blood pressure <135/80 mmHg | 74.3
  Blood pressure <130/80 mmHg | 69.9
  Blood pressure <120/80 mmHg | 43.4

58. Secondary Outcome: Percentage of Participants Previously on a Nondihydropyridine Calcium Channel Blocker Achieving the Blood Pressure Goals From Baseline to 12 Weeks
Time Frame: Baseline to 12 weeks
Population: Participants previously on a Nondihydropyridine Calcium Channel Blocker who have received at least one dose of study medication and who have a baseline value.
Measure: Number; unit: Percentage of participants
Arm/Group | Olmesartan Medoxomil/Amlodipine Tablets + Hydrochlorothiazide
Number analyzed (Participants) | 20
Percentage of participants
  Systolic blood pressure <140 mmHg | 100.0
  Systolic blood pressure <135 mmHg | 90.0
  Systolic blood pressure <130 mmHg | 75.0
  Systolic blood pressure <120 mmHg | 25.0
  Diastolic blood pressure <90 mmHg | 100.0
  Diastolic blood pressure <85 mmHg | 95.0
  Diastolic blood pressure <80 mmHg | 75.0
  Blood pressure <140/90 mmHg | 100.0
  Blood pressure <135/80 mmHg | 70.0
  Blood pressure <130/80 mmHg | 65.0
  Blood pressure <120/80 mmHg | 20.0

59. Secondary Outcome: Percentage of Participants Previously on a Nondihydropyridine Calcium Channel Blocker Achieving the Blood Pressure Goals From Baseline to 20 Weeks
Time Frame: Baseline to 20 weeks
Population: as for outcome 58
Measure: Number; unit: Percentage of participants
Arm/Group | Olmesartan Medoxomil/Amlodipine Tablets + Hydrochlorothiazide
Number analyzed (Participants) | 20
Percentage of participants
  Systolic blood pressure <140 mmHg | 100.0
  Systolic blood pressure <135 mmHg | 100.0
  Systolic blood pressure <130 mmHg | 95.0
  Systolic blood pressure <120 mmHg | 45.0
  Diastolic blood pressure <90 mmHg | 100.0
  Diastolic blood pressure <85 mmHg | 95.0
  Diastolic blood pressure <80 mmHg | 95.0
  Blood pressure <140/90 mmHg | 100.0
  Blood pressure <135/80 mmHg | 95.0
  Blood pressure <130/80 mmHg | 95.0
  Blood pressure <120/80 mmHg | 40.0

ADVERSE EVENTS:
Time Frame: Adverse events were collected for the 20-week treatment period + a 2-week post-treatment follow-up, plus an additional 30 days after last dose.
Description: AE's were either observed by the investigator via physical examinations and laboratory testing and/or reported by the subject.
Arm/Group | Olmesartan Medoxomil/Amlodipine Tablets + Hydrochlorothiazide
Serious Adverse Events (participants affected / at risk) | 13/999
Other Adverse Events (participants affected / at risk) | 241/999
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Olmesartan Medoxomil/Amlodipine Tablets + Hydrochlorothiazide (N=999)
myocardial infarction (Cardiac disorders) | 2 (2)
depession (Psychiatric disorders) | 1 (1)
oesophageal rupture (Gastrointestinal disorders) | 1 (1)
presyncope (Nervous system disorders) | 1 (1)
epilepsy (Nervous system disorders) | 1 (1)
Non small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
abdominal pain (Gastrointestinal disorders) | 1 (1)
vaginal haemhorrage (Reproductive system and breast disorders) | 1 (1)
road traffic accident (Injury, poisoning and procedural complications) | 1 (1)
muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
protate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2.0% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Olmesartan Medoxomil/Amlodipine Tablets + Hydrochlorothiazide (N=999)
oedema (General disorders) | 86
headache (Nervous system disorders) | 52
dizziness (Nervous system disorders) | 103

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
As stated in the clinical study agreement, If identified by DSI, any of DSI's confidential information as defined herein shall be deleted...Nothing in this publication section shall be taken as giving DSI any right of editorial control over any publicartion prepared by the Study Site."